# ECOPIPAM (EBS-101) EBS-101-OL-001

**IND Number:** 109746

**EudraCT Number:** 2019-000282-20

**Protocol Title:** A Multicenter, Open-Label, Extension Study Intended to

Evaluate the Long-term Safety of Ecopipam Tablets in Children and Adolescent Subjects with Tourette's

Syndrome

**Indication Studied:** Children and Adolescent Subjects with Tourette's Syndrome

**Protocol Version/Date:** 7.0, Amendment 6, 17 November 2021

**Sponsor Address:** Emalex Biosciences, Inc.

300 North Wabash Avenue, Suite 3500

Chicago, IL, 60611

The program will be completed according to the guidelines of Good Clinical Practice. Compliance with this standard provides public assurance that the rights, safety, and well-being of trial subjects are protected, consistent with the principles that have their origin in the Declaration of Helsinki.

#### **Confidentiality Statement**

The information in this document contains trade and commercial information that is privileged or confidential and may not be disclosed unless such disclosure is required by federal or state law or regulations. In any event, persons to whom the information is disclosed must be informed that the information is privileged or confidential and may not be further disclosed by them. These restrictions on disclosure will apply equally to all future information supplied to you which is indicated as privileged or confidential.

# 1. PROTOCOL AMENDMENT CHANGES

 Table 2:
 Study Design and Schedule of Assessments

# **Existing Text**

| Assessment <sup>4</sup> | Baseline*<br>(Titration) | | | | | Tr | eatm | ent | | | | | End of Study<br>/ Early<br>Termination | Follow Up<br>Visit | Follow Up<br>Phone Call |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Month | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | One and<br>Two Weeks<br>Post Last<br>Dose | 30 Days<br>After Last<br>Dose |
| Study Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 & 15 | |
| Visit Window | | ±3<br>days | ±3<br>days | ±3<br>days | ±3<br>days | ±3<br>days | ±3<br>days | ±3<br>days | ±3<br>days | ±3<br>days | ±3<br>days | ±3 | ±3 <sub>days</sub> | ±3 <sub>days</sub> | ±3 <sub>days</sub> |
| Informed Consent | X | | | | | | | | | | | | | | |
| Inclusion/ Exclusion | X | | | | | | | | | | | | | | |
| Medical/Psychiatric/<br>Medication History | X | | | | | | | | | | | | | | |
| Physical Examination | X | X | | X | | | X | | | X | | | X | X | |
| Vital Signs <sup>1</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| ECG | X | X | | X | | | X | | | X | | | X | | |
| Laboratory Tests<br>(Hematology and<br>Chemistry) <sup>2</sup> | X | X | | X | | | X | | | X | | | X | X | |
| Urine Drug Screen | X | X | | X | | | X | | | X | | | X | | |
| Urine Pregnancy Test | X | X | | X | | | X | | | X | | | X | | |


| Assessment <sup>4</sup> | Baseline* (Titration) | | | | | Tr | eatm | ent | | | | | End of Study<br>/ Early<br>Termination | Follow Up<br>Visit | Follow Up<br>Phone Call |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Month | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | One and<br>Two Weeks<br>Post Last<br>Dose | 30 Days<br>After Last<br>Dose |
| Study Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 & 15 | |
| HbA1c | | X | | X | | | X | | | X | | | X | | |
| YGTSS Score | X | X | | X | | | X | | | X | | | X | | |
| CGI-TS-I | | X | | X | | | X | | | X | | | X | | |
| CGI-TS-S | X | X | | X | | | X | | | X | | | X | | |
| C&A-GTS-QOL | X | X | | X | | | X | | | X | | | X | | |
| Columbia Suicide<br>Severity Rating Scale | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Abnormal Involuntary<br>Movement Scale<br>(AIMS) | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Barnes Akathisia<br>Ratings Scale (BARS) | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Children's Depression<br>Rating Scale-Revised<br>(CDRS-R) | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Pediatric Anxiety<br>Ratings Scale (PARS) | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Adverse Events | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant<br>Medications | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |


| Assessment <sup>4</sup> | Baseline*<br>(Titration) | | | | | Tr | eatmo | ent | | | | | End of Study<br>/ Early<br>Termination | Follow Up<br>Visit | Follow Up<br>Phone Call |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Month | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | One and<br>Two Weeks<br>Post Last<br>Dose | 30 Days<br>After Last<br>Dose |
| Study Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 & 15 | |
| Dispense Study Drug | X | X | X | X | X | X | X | X | X | X | X | X | $X^3$ | | |
| Collect Unused Study<br>Drug/Assess Drug<br>Compliance | | X | X | X | X | X | X | X | X | X | X | X | X | X | |

Abbreviations: BP = blood pressure, CGI = Clinician Global Impression, CGI-TS-I = CGI Tourette Syndrome of Improvement, CGI-TS-S = CGI Tourette Syndrome of Severity, ECG = electrocardiogram, HbA1c = Hemoglobin A1c


<sup>\*</sup> Baseline is to occur within 30 days of the EBS-101-CL-001 14 Day Follow Up Visit (or longer with the permission of the medical monitor). All Baseline measurements can be taken from the Day 14 Follow Up Visit of the EBS-101-CL-001 study if performed less than 7 days prior to the Baseline visit. In this case, the HbA1c and Urine Drug Screen from the Week 12/Completion Visit of the EBS-101-CL-001 study may be used.

<sup>&</sup>lt;sup>1</sup> Vital signs will include heart rate, BP, orthostatic BP and heart rate (done supine and then 3 minutes after standing), height and weight.

<sup>&</sup>lt;sup>2</sup> Subjects should be in a fasting state (8 hours) for laboratory tests.

<sup>&</sup>lt;sup>3</sup> Study drug dispensation for down titration.

<sup>&</sup>lt;sup>4</sup> Assessments for Study Visits may be completed in locations other than study clinic and/or safety and efficacy assessments required at these visits will be made available for remote administration due to restrictions as a consequence of the COVID-19 pandemic or other qualifying event.

# **Revised Text**

| Assessment <sup>4</sup> | Baseline* (Titration) | | | | | Tr | eatmo | ent | | | | | End of Study<br>/ Early<br>Termination | Follow Up<br>Visit | Follow Up<br>Phone Call |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Month | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | One and<br>Two Weeks<br>Post Last<br>Dose | 30 Days<br>After Last<br>Dose |
| Study Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 & 15 | |
| Visit Window | | ±3<br>days | ±3 | ±3<br>days | ±3 | ±3 | ±3 | ±3<br>days | ±3<br>days | ±3<br>days | ±3 | ±3<br>days | ±3 <sub>days</sub> | ±3days | $\pm 3$ days |
| Informed Consent | X | | | | | | | | | | | | | | |
| Inclusion/ Exclusion | X | | | | | | | | | | | | | | |
| Medical/Psychiatric/<br>Medication History | X | | | | | | | | | | | | | | |
| Physical Examination | X | X | | X | | | X | | | X | | | X | X | |
| Vital Signs <sup>1</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| ECG | X | X | | X | | | X | | | X | | | X | | |
| Laboratory Tests<br>(Hematology,<br>Chemistry and<br>Urinalysis) <sup>2</sup> | X | X | | X | | | X | | | X | | | X | X | |
| Urine Drug Screen | X | X | | X | | | X | | | X | | | X | | |
| Urine Pregnancy Test | X | X | | X | | | X | | | X | | | X | | |
| HbA1c | | X | | X | | | X | | | X | | | X | | |
| YGTSS Score | X | X | | X | | | X | | | X | | | X | | |
| CGI-TS-I | | X | | X | | | X | | | X | | | X | | |


| Assessment <sup>4</sup> | Baseline* (Titration) | | | | | Tr | eatm | ent | | | | | End of Study<br>/ Early<br>Termination | Follow Up<br>Visit | Follow Up<br>Phone Call |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Month | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | One and<br>Two Weeks<br>Post Last<br>Dose | 30 Days<br>After Last<br>Dose |
| Study Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 & 15 | |
| CGI-TS-S | X | X | | X | | | X | | | X | | | X | | |
| C&A-GTS-QOL | X | X | | X | | | X | | | X | | | X | | |
| Columbia Suicide<br>Severity Rating Scale | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Abnormal Involuntary<br>Movement Scale<br>(AIMS) | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Barnes Akathisia<br>Ratings Scale (BARS) | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Children's Depression<br>Rating Scale-Revised<br>(CDRS-R) | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Pediatric Anxiety<br>Ratings Scale (PARS) | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Adverse Events | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant<br>Medications | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Dispense Study Drug | X | X | X | X | X | X | X | X | X | X | X | X | $X^3$ | | |
| Collect Unused Study<br>Drug/Assess Drug<br>Compliance | | X | X | X | X | X | X | X | X | X | X | X | X | X | |


Abbreviations: BP = blood pressure, CGI = Clinician Global Impression, CGI-TS-I = CGI Tourette Syndrome of Improvement, CGI-TS-S = CGI Tourette Syndrome of Severity, ECG = electrocardiogram, HbA1c = Hemoglobin A1c

- \* Baseline is to occur within 30 days of the EBS-101-CL-001 14 Day Follow Up Visit (or longer with the permission of the medical monitor). All Baseline measurements can be taken from the Day 14 Follow Up Visit of the EBS-101-CL-001 study if performed less than 7 days prior to the Baseline visit. In this case, the HbA1c and Urine Drug Screen from the Week 12/Completion Visit of the EBS-101-CL-001 study may be used.
- <sup>1</sup> Vital signs will include heart rate, BP, orthostatic BP and heart rate (done supine and then 3 minutes after standing), height and weight.
- <sup>2</sup> Subjects should be in a fasting state (8 hours) for laboratory tests.
- <sup>3</sup> Study drug dispensation for down titration.
- <sup>4</sup> Assessments for Study Visits may be completed in locations other than study clinic and/or safety and efficacy assessments required at these visits will be made available for remote administration due to restrictions as a consequence of the COVID-19 pandemic or other qualifying event.

#### **Rationale for Amendment**

Urinalysis is being added.

**Section: 12.1 Safety Parameters** 

**Existing Text** 

**Clinical Laboratory Tests** 

<u>Category</u> <u>Parameters</u>

Hematology Red blood cell count, hemoglobin,

hematocrit, platelets, and white blood cell count with differential (neutrophils, bands lymphocytes, monocytes, eosinophils,

basophils)

Chemistry

Electrolytes Sodium, potassium, chloride, bicarbonate

Liver function tests Alkaline phosphatase, aspartate

aminotransferase (AST), alanine

aminotransferase (ALT), total bilirubin,

direct bilirubin

Renal function parameters Blood urea/blood urea nitrogen (BUN),

creatinine

Other Glucose, calcium, albumin, cholesterol,

triglycerides, phosphorus, lactate dehydrogenase (LDH), total protein,

globulin

Pregnancy Test Urine test (for women of childbearing

potential only)

**Special Parameters - Hemoglobin** 

**A1c** (HbA1c)

#### **Revised Text**

## **Clinical Laboratory Tests**

<u>Category</u> <u>Parameters</u>

Hematology Red blood cell count, hemoglobin,

hematocrit, platelets, and white blood cell count with differential (neutrophils, bands lymphocytes, monocytes, eosinophils,

basophils)

Chemistry

Electrolytes Sodium, potassium, chloride, bicarbonate

Liver function tests Alkaline phosphatase, aspartate

aminotransferase (AST), alanine

aminotransferase (ALT), total bilirubin,

direct bilirubin

Renal function parameters Blood urea/blood urea nitrogen (BUN),

creatinine

| Emalex Biosciences, Inc. | Protocol EBS-101-OL-001 |
|--------------------------|--------------------------------------------|
| Ecopipam | Version 7.0, Amendment 6, 17 November 2021 |

Other Glucose, calcium, albumin, cholesterol,

triglycerides, phosphorus, lactate dehydrogenase (LDH), total protein,

globulin

Urinalysis Complete urinalysis includes color,

appearance, specific gravity, pH, protein,

glucose, ketones, and blood with microscopic examination for positive

protein or blood results

Urine test (for women of childbearing

potential only)

**Pregnancy Test** 

**Special Parameters - Hemoglobin** 

A1c (HbA1c)

### **Rationale for Amendment**

Urinalysis is being added.

#### **SIGNATURE PAGE**

## Sponsor's Approval

The protocol has been approved by Emalex Biosciences, Inc.

This program will be conducted with the highest respect for the individual participants in accordance with the requirements of this clinical protocol and also in accordance with the following:

- The ethical principles that have their origin in the Declaration of Helsinki.
- International Conference on Harmonization (ICH) Tripartite: Harmonized Guideline for Good Clinical Practice E6.
- All applicable laws and regulations, including, without limitation, data privacy laws and regulations.



# INVESTIGATOR'S AGREEMENT

| I have received and read the Investigator's Brochure for Ecopipam. I have read the protocol EBS-101-OL-001 and agree to conduct the study as outlined. I agree to maintain the confidentiality of all information received or developed in connection with this protocol. |
|---|
| Printed Name of Investigator |
| Signature of Investigator |
| Date |

# PROCEDURES IN CASE OF EMERGENCY

**Table 1:** Emergency Contact Information

| Role in Study | Name | Contact Information |
|---------------------------|--------------------------|---------------------|
| Clinical Study Leader | PPD | PPD |
| | | PPD |
| Drug Safety Physician | Syneos Medical Physician | 1 877-462-0134 |
| 24-Hour emergency contact | Syneos Medical Physician | 1 877-462-0134 |

### 2. SYNOPSIS

#### Name of Sponsor/Company:

Emalex Biosciences, Inc.

#### Name of Investigational Product:

**Ecopipam Tablets** 

Protocol Number: EBS-101-OL-001

#### **Title of Study:**

A Multicenter, Open-Label, Extension Study Intended to Evaluate the Long-term Safety of Ecopipam Tablets in Children and Adolescent Subjects with Tourette's Syndrome

Study center(s): Approximately 60 sites in US, Canada and EU

**Principal Investigator:** TBD

**Investigators:** TBD

#### Studied period (years):

Estimated date first patient enrolled: 3Q2019

Estimated date last patient completed: 2Q2023, or until NDA

approval or until development is discontinued by the

Sponsor, whichever is sooner

#### **Phase of development:**

2b

### **Objectives:**

The primary objective of this study is to evaluate the long-term safety and tolerability of ecopipam tablets in pediatric subjects (aged  $\geq 6$  to  $\leq 18$  years at Baseline) with Tourette's Syndrome (TS) that were previously enrolled in the EBS-101-CL-001 study (Phase 2b) and completed the Phase 2b study. The secondary objective is to evaluate the durability of effect of ecopipam in pediatric subjects (aged  $\geq 6$  to  $\leq 18$  years at Baseline) with TS.

#### Methodology:

This is an international, multicenter, open-label, long-term extension study evaluating the safety of ecopipam tablets for the treatment of children and adolescent subjects with TS. Subjects who completed the Phase 2b, randomized double-blind efficacy and safety study (EBS-101-CL-001) and who continue to meet the inclusion/exclusion criteria for this study will be eligible to participate in this study. All subjects will be titrated to a target dose of 2 mg/kg/day as subjects participating from previous studies will be tapered off of study medication to maintain the blind. Subjects will complete study visits every month for 1 year. Follow Up visits will be conducted 7 and 14 days after the last dose of study medication and a Follow Up phone call will be conducted 30 days after the last dose of study medication. Study Visits may be completed in locations other than clinic and/or safety and efficacy assessments required at these visits will be made available for remote administration due to restrictions as a consequence of the COVID-19 pandemic or other qualifying event.

Safety will be monitored throughout the study at all visits by repeated adverse event (AE) monitoring, vital signs, the Columbia-Suicide Severity Rating Scale (C-SSRS), the Abnormal Involuntary Movement Scale (AIMS), the Barnes Akathisia Rating Scale (BARS), the Pediatric Anxiety Rating Scale (PARS) and Children's Depression Rating Scale-Revised (CDRS-R). In addition to these assessments, at Baseline, Months 1, 3, 6, 9 and 12 safety will also be monitored by clinical and laboratory evaluations, and electrocardiogram (ECG) monitoring. In addition to the scales aforementioned, the Yale Global Tic Severity Scale (YGTSS), Clinician Global Impression of Tourette Syndrome of Severity (CGI-TS-S), the Clinician Global Impression Tourette Syndrome of

Improvement (CGI-TS-I) and the Gilles de la Tourette Syndrome—Quality of Life Scale for Children and Adolescents (C&A-GTS-QOL) will also be assessed at Baseline, Months 1, 3, 6, 9 and 12. At the Follow Up visits, AE monitoring, the C-SSRS, clinical and laboratory evaluations and vital signs will be assessed. A Follow Up phone call will be conducted 30 days after the last dose of study medication to assess AEs.

#### Number of subjects (planned):

The actual number of subjects that are enrolled will depend on the final number of subjects who complete the Phase 2b, randomized double-blind efficacy and safety study (EBS-101-CL-001) and who continued to meet the inclusion and exclusion criteria for this study.

#### Diagnosis and main criteria for inclusion:

#### Inclusion Criteria:

- 1) Subjects must have completed the EBS-101-CL-001 study through the Day 14 Follow Up Visit within the last 30 days (or longer with permission of the medical monitor) and must be who the Investigator feels would benefit from continued participation.
- 2) Adolescent females of childbearing potential who are sexually active must be using highly effective contraception (i.e., oral contraceptives, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomized male partner) and agree to continue use of highly effective contraception for the duration of their participation in the study. They must also agree to use highly effective contraception for 30 days after their last dose of study drug.
- 3) Sexually active male subjects must use a highly effective method of contraception during the study and agree to continue the use of highly effective contraception for at least 30 days after the last dose of study drug.
- 4) Parents or legal guardians of subjects <18 years of age at Baseline must execute a written informed consent. Subjects ≥18 years of age must execute a written informed consent.
- 5) Subjects <18 years of age at Baseline must execute a written informed assent according to the requirements of the site's IRB/EC.

#### Exclusion Criteria:

- 1) Subjects with a clinical presentation and/or history consistent with another neurologic condition that may have had accompanying abnormal movements (e.g., Huntington's disease, Parkinson's disease, Wilson's disease, stroke, Restless Legs Syndrome).
- 2) History of schizophrenia, bipolar disorder, or other psychotic disorders.
- 3) Any unstable primary mood disorder (DSM-5 criteria) at time of Baseline.
- 4) Subjects who have unstable medical illness or clinically significant abnormalities on laboratory tests or ECG at Baseline as determined by the Principal Investigator.
- 5) Subjects who have moderate to severe renal insufficiency at Screening.
- 6) Subjects with a major depressive episode in the past 2 years.
- 7) Subjects with a history of attempted suicide.
- 8) A significant risk of committing suicide based on history, routine psychiatric status examination, Investigator's judgment, or who had an answer of "yes" on any question other than 1–3 (currently or within the past 30 days) on the baseline/screening version of the C-SSRS.
- 9) Subjects with a history of seizures (excluding febrile seizures that occurred <2 years prior to Baseline).
- 10) Subjects with a myocardial infarction within 6 months.
- 11) Female subjects who are currently pregnant or lactating or planning to get pregnant during the course of the study.

- 12) Subjects who have a need for medications which would have unfavorable interactions with ecopipam, e.g., dopamine antagonists or agonists [including bupropion], tetrabenazine, monoamine oxidase inhibitors, or St. John's Wort.
- 13) Subjects with current or recent (past 3 months) DSM-5 substance use disorder (with the exception of nicotine).
- 14) Subjects with positive urine drug screen for cocaine, amphetamine, methamphetamine, benzodiazepines, barbiturates, phencyclidine (PCP) or opiates at Baseline, except those receiving stable, prescribed treatment for attention deficit/hyperactivity disorder. Subjects with urine positive only for benzodiazepines will be exclusionary unless medically prescribed.
- 15) Subjects with a lifetime history of bipolar disorder type I or II, dementia, schizophrenia, or any other psychotic disorder.
- 16) Inability to swallow tablets.
- 17) Subjects with a known hypersensitivity to ecopipam or any of its excipients.
- 18) Any subject who in the opinion of the investigator is not a suitable candidate for the study.

## Investigational product, dosage and mode of administration:

Ecopipam HCl will be supplied as 12.5-, 37.5-, 50-, 75-, and 100-mg tablets. The target dose is 2 mg/kg via oral administration.

Subjects will be dosed according to the following weight bands to better achieve the 2 mg/kg/day target dose:  $\geq 18-\leq 23$  kg,  $\geq 23-\leq 34$  kg,  $\geq 34-\leq 44$  kg,  $\geq 44-\leq 68$  kg,  $\geq 68-\leq 83$  kg,  $\geq 83$  kg.

During the 4-week titration period, the following ecopipam HCl doses will be administered for each of the weight bands:

- Those who weigh ≥18-≤23 kg will titrate from 12.5 mg daily to 37.5 mg daily: 12.5 mg during Week 1, 25 mg during Week 2, and 37.5 mg during Weeks 3 and 4.
- Those who weigh >23-\le 34 kg will titrate from 12.5 mg daily to 50 mg daily: 12.5 mg during Week 1, 25 mg during Week 2, 37.5 mg during Week 3, and 50 mg during Week 4.
- Those who weigh >34- $\leq$ 44 kg will titrate from 12.5 mg daily to 75 mg daily: 12.5 mg during Week 1, 25 mg during Week 2, 50 mg during Week 3, and 75 mg during Week 4.
- Those who weigh >44-≤68 will titrate from 25 mg daily to 100 mg daily: 25 mg during Week 1, 50 mg during Week 2, 75 mg during Week 3, and 100 mg during Week 4.
- Those who weigh >68- $\leq$ 83 kg will titrate from 25 mg daily to 150 mg daily: 25 mg during Week 1, 50 mg during Week 2, 100 mg during Week 3, and 150 mg during Week 4.
- Those who weigh >83 kg will titrate from 25 mg daily to 200 mg daily: 25 mg during Week 1, 50 mg during Week 2, 100 mg during Week 3, and 200 mg during Week 4.

During the 52-week treatment phase, the following ecopipam doses will be administered for each of the weight bands:

- Those who weigh  $\ge 18 \le 23$  kg will receive 37.5 mg daily.
- Those who weigh >23-\le 34 kg will receive 50 mg daily.
- Those who weigh >34-≤44 will receive 75 mg daily.
- Those who weigh >44-≤68 kg will receive 100 mg daily.
- Those who weigh >68-\le 83 kg will receive 150 mg daily.
- Those who weigh >83 kg will receive 200 mg daily.

At the end of the 52-week treatment phase, subjects will titrate off therapy and receive ecopipam HCl doses that will be reduced by 25 mg/day until off drug.

#### **Duration of treatment:**

52-weeks, until New Drug Application (NDA) approval, or until development of the study drug is discontinued by the Sponsor, whichever is sooner.

#### **Criteria for evaluation:**

**Safety:** Study Visits may be completed in locations other than clinic and/or safety and efficacy assessments required at these visits will be made available for remote administration due to restrictions as a consequence of the COVID-19 pandemic or other qualifying event. Safety will be monitored throughout the study at every visit by repeated adverse event (AE) monitoring, vital signs, the Columbia-Suicide Severity Rating Scale (C-SSRS), the Abnormal Involuntary Movement Scale (AIMS), the Barnes Akathisia Rating Scale (BARS), the Pediatric Anxiety Rating Scale (PARS) and Children's Depression Rating Scale-Revised (CDRS-R). In addition to these assessments, at Baseline, Months 1, 3, 6, 9 and 12 safety will also be monitored by clinical and laboratory evaluations and electrocardiogram (ECG) monitoring. At the Follow Up visits, AE monitoring, the C-SSRS, clinical and laboratory evaluations and vital signs will be assessed. Laboratory evaluations will include hematology, chemistry, urine values and HbA1c. A Follow Up phone call will be conducted 30 days after the last dose of study medication to assess AEs. Subjects will be monitored for signs of abuse, and withdrawal or dependence.

**Efficacy:** The YGTSS, CGI-TS-S and C&A-GTS-QOL will be conducted at Baseline and Months 1, 3, 6, 9 and 12. The CGI-TS-I will be conducted at Months 1, 3, 6, 9, and 12.

All safety and efficacy variables will be summarized descriptively.

Additional analyses may need to be conducted for data not collected at sites and/or collected via remote administration due to restrictions as a consequence of the COVID-19 pandemic or other qualifying event, these additional analyses will be specified in the SAP.

| 3 | • | <b>TABLE</b> | OF | CON | TENTS |
|---|---|--------------|----|-----|-------|
|---|---|--------------|----|-----|-------|

| 1. | PROTOCOL AMENDMENT CHANGES | 2 |
|----------|---------------------------------------------------|----|
| SIGNATU | RE PAGE | 10 |
| INVESTIG | GATOR'S AGREEMENT | 11 |
| PROCEDU | JRES IN CASE OF EMERGENCY | 12 |
| 2. | SYNOPSIS | 13 |
| 3. | TABLE OF CONTENTS | 17 |
| 4. | LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 20 |
| 5. | INTRODUCTION | 21 |
| 5.1. | Background on Tourette's Syndrome | 21 |
| 5.1.1. | Disrupted Dopamine Systems in Tourette's Syndrome | 22 |
| 5.2. | Background on Ecopipam. | 23 |
| Cl | | |
| 5.2.2. | Clinical Data | 23 |
| 5.2.2.1. | Safety in Humans | 23 |
| 5.3. | Risk-Benefit Assessment | 27 |
| 5.3.1. | Assessment of Risk | 27 |
| 5.3.2. | Assessment of Benefit | 28 |
| 5.3.3. | Methods to Minimize Risks | 29 |
| 6. | STUDY OBJECTIVES AND PURPOSE | 31 |
| 6.1. | Primary Objective | 31 |
| 6.2. | Secondary Objectives | 31 |
| 7. | INVESTIGATIONAL PLAN | 32 |
| 7.1. | Overall Study Design. | 32 |
| 7.2. | Number of Subjects | 32 |
| 7.3. | Treatment Assignment | 32 |
| 7.4. | Dose Adjustment Criteria | 32 |
| 7.5. | Criteria for Subject Study Discontinuation | 33 |
| 8. | SELECTION AND WITHDRAWAL OF SUBJECTS | 37 |
| 8.1. | Subject Inclusion Criteria | 37 |
| 8.2. | Subject Exclusion Criteria | 37 |
| 8.3. | Subject Withdrawal Criteria | 38 |

| 9. | TREATMENT OF SUBJECTS | 39 |
|-----------|-------------------------------------|----|
| 9.1. | Description of Study Drug | 39 |
| 9.2. | Concomitant Medications | 39 |
| 9.3. | Prohibited Therapies | 39 |
| 9.4. | Treatment Compliance | 40 |
| 9.5. | Randomization and Blinding | 40 |
| 10. | STUDY DRUG MATERIALS AND MANAGEMENT | 41 |
| 10.1. | Study Drug | 41 |
| 10.2. | Study Drug Packaging and Labeling | 41 |
| 10.3. | Study Drug Storage | 41 |
| 10.4. | Study Drug Preparation | 41 |
| 10.5. | Administration | 41 |
| 10.6. | Dosing Rationale | 43 |
| 10.7. | Study Drug Accountability | 45 |
| 10.8. | Study Drug Handling and Disposal | 45 |
| 11. | ASSESSMENT OF EFFICACY | 46 |
| 11.1 | Efficacy Assessments | 46 |
| 12. | ASSESSMENT OF SAFETY | 47 |
| 12.1. | Safety Parameters | 47 |
| 12.2. | Adverse and Serious Adverse Events | 48 |
| 12.2.1. | Definition of Adverse Events | 48 |
| 12.2.1.1. | Treatment-Emergent Adverse Event | 49 |
| 12.2.1.2. | Serious Adverse Event | 49 |
| 12.2.1.3. | Other Adverse Event | 49 |
| 12.3. | Relationship to Study Drug | 50 |
| 12.4. | Recording Adverse Events | 50 |
| 12.5. | Reporting Adverse Events | 51 |
| 13. | STATISTICS | 52 |
| 13.1. | Analysis Populations | 52 |
| 13.2. | Planned Analyses | 52 |
| 13.2.1. | Safety Analysis | 52 |
| 13.2.2. | Efficacy Analysis | 53 |

| E : |
|----------|
| Ecopipam |

| 14. | DIRECT ACCESS TO SOURCE DATA/DOCUMENTS | 54 |
|---|---|---|
| 14.1. | Study Monitoring | 54 |
| 14.2. | Audits and Inspections | 54 |
| 14.3. | Institutional Review Board (IRB)/Independent Ethics Committee (IEC) | 55 |
| 15. | QUALITY CONTROL AND QUALITY ASSURANCE | 56 |
| 16. | ETHICS | 57 |
| 16.1. | Ethics Review | 57 |
| 16.2. | Ethical Conduct of the Study | 57 |
| 16.3. | Written Informed Consent | 57 |
| 16.4. | Subject Confidentiality | 57 |
| 17. | DATA HANDLING AND RECORDKEEPING | 59 |
| 17.1. | Inspection of Records | 59 |
| 17.2. | Retention of Records | 59 |
| 18. | PUBLICATION POLICY | 60 |
| 19. | LIST OF REFERENCES | 61 |
| 20. | REFERENCES FOR QUESTIONNAIRES AND SCALES | 62 |
| 21. | APPENDICES | 63 |
| WMA DE | ECLARATION OF HELSINKI – ETHICAL PRINCIPLES FOR MEDICAL RESEARCH INVOLVING HUMAN SUBJECTS | 63 |
| CONTRA | CEPTION GUIDELINES | 69 |
| PROHIBI | TED MEDICATIONS LIST | 70 |
| | LIST OF TABLES | |
| Table 1: | Emergency Contact Information | 12 |
| Table 2: | Study Design and Schedule of Assessments | 34 |
| Table 3: | Investigational Product | 39 |
| Table 4: | Proposed Dosing Regimen | 43 |
| Table 5: | Animal:Human Exposure Ratios with the Proposed Dosage Regimen of Ecopipam HCl to 7 to 16 Year Olds | 44 |

# 4. LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

The following abbreviations and specialist terms are used in this study protocol.

| Abbreviations | Terms |
|---|---|
| ADD | attention deficit disorder |
| ADHD | attention deficit/hyperactivity disorder |
| AE | adverse event |
| AESI | adverse event of special interest |
| AIMS | Abnormal Involuntary Movement Scale |
| CDRS-R | Children's Depression Rating Scale-Revised |
| CGI | Clinician Global Impression |
| CGI-TS-I | Clinician Global Impression Tourette's Syndrome of Improvement |
| CGI-TS-S | Clinician Global Impression Tourette's Syndrome of Severity |
| CI | confidence interval |
| COVID-19 | SARS-CoV-2 (coronavirus) |
| CRF | case report form |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| CY-BOCS | Child Yale-Brown Obsessive Compulsive |
| DSM-5 | Diagnostic and Statistical Manual of Mental Disorders – 5th |
| | Edition |
| ECG | electrocardiogram |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practices |
| HC1 | Hydrochloride |
| HbA1c | Hemoglobin A1c |
| ITT | Intent-to-treat |
| ICH | International Conference on Harmonisation of Technical Requirements |
| | for Registration of Pharmaceuticals for Human Use |
| IEC | Independent Ethics Committee |
| IRB | Institutional Review Board |
| LND | Lesch-Nyhan Disease |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mITT | modified intent-to-treat |
| OAE | other adverse event |
| OCD | obsessive-compulsive disorder |
| PARS | Pediatric Anxiety Rating Scale |
| PO | oral (per os) |
| SAE | serious adverse event |
| SCH | Schering-Plough drug code indicator |
| SD | standard deviation |
| TEAE | treatment-emergent adverse event |
| TS | Tourette's Syndrome |
| US | United States |
| YGTSS | Yale Global Tic Severity Score |

### 5. INTRODUCTION

## 5.1. Background on Tourette's Syndrome

Tourette's Syndrome (TS) is a neurological disorder characterized by motor or vocal tics that begin in childhood and persist over time (see box below with the Diagnostic and Statistical Manual for Mental Disorders – 5th Edition [DSM-5] diagnostic criteria). The tics are brief in duration, occur spontaneously, and do not show a regular temporal pattern. Further, the tics are not caused by medications, other medical reasons, or confirmed neurological abnormality. They can be consciously suppressed for some time and are exacerbated by stress. Males are more susceptible than females, with a ratio of about 4.1 to 3. Motor tics can include such things as eye-blinking, facial grimacing, mouth movements, head jerks, shoulder shrugs, and arm/leg jerks. In more severe cases, gyrating, bending, pivoting, and dystonic movements are possible. Vocal tics are fast meaningless sounds or noises, and include such things as sniffing, throat clearing, grunting, barks, and squealing. Complex vocal tics can include shouting out of single words, whole sentences or repeating words (echolalia). In small numbers of subjects, explosive obscenities (coprolalia) are possible. 1.2 Diagnosis of TS is complicated because it often co-exists with other psychiatric illnesses. Common co-morbid conditions include attention deficit/hyperactivity disorder (ADHD), obsessive-compulsive disorder (OCD), anxiety, and depression.<sup>2</sup> These symptoms often mask TS and make diagnosis difficult. Tic severity can range from mild to severe according to its frequency and intensity. The tics have a variable course, with severe bouts interspersed with complete absence of symptoms. Onset of tics is seen early in childhood (average approximately 7 years) and peaks in the teenage years. Vocal tics appear several years after the onset of motor tics. For most subjects, the period of worst-ever tic severity is between 7 and 15 years old, followed by a steady decline in tic severity. As subjects mature, the vast majority of tics will disappear permanently, with a small percentage of subjects having tics that persist into adulthood and require treatment. Complete remission of tics is reported in approximately 50% of subjects. Severe tics are thought to occur only in about 10% of the cases. $\frac{3}{2}$ 

## DSM-V Diagnostic Criteria For Tourette's Syndrome

**Note:** A *tic* is a sudden, rapid, recurrent, nonrhythmic, stereotyped motor movement or vocalization.

- A. Both multiple motor and one or more vocal tics have been present at some time during the illness, although not necessarily concurrently.
- B. The tics may wax and wane in frequency but have persisted for more than 1 year since first tic onset.
- C. The onset is before age 18 years.
- D. The disturbance is not attributable to the physiological effects of a substance (e.g. Cocaine) or another medical condition (e.g. Huntington's disease, postviral encephalitis).

## Natural History of Tics



Approaches to the treatment of tics include: education, behavioral therapy, pharmacological therapy, and treatment of comorbid conditions (attention deficit disorder [ADD], OCD). Approximately, 20% of subjects do not need treatment. Counseling and behavioral therapy may be sufficient with mild symptoms. Medications should be considered when tics interfere with peer relationships, social interactions, job or school performance, or activities of daily living. Medications should be started at low doses, titrated up slowly to lowest effective dose, and tapered slowly during non-stressful periods. Medication therapy incudes: dopamine receptor blocking agents, dopamine depleting agents, benzodiazepines, low dose dopamine agonists, botulinum toxin, and neurosurgical treatment. Non-selective dopamine receptor blocking agents have been the mainstay of treatment and are the most effective. They suppress tics in 70-80% of patients. Many patients eventually discontinue due to adverse events (AEs), including extrapyramidal disorders, somnolence, blood glucose changes, weight gain, and effects on lipids. A selective D1 dopamine receptor blocking agent may mitigate against some of these AEs and has the potential to offer a safer alternative option.

### 5.1.1. Disrupted Dopamine Systems in Tourette's Syndrome

The underlying mechanism responsible for TS is unknown. Although the disease tends to run in families, there have been no definitive genetic mutations identified.<sup>4</sup> Research to date has indicated that dopamine circuits in the central nervous system (CNS) are intimately involved based on the following observations.<sup>5,6,7</sup>

- Dopamine-rich areas of the brain (e.g., striatum) are believed to control motor tics.
- Clinical neuroimaging studies of TS patients implicate dopamine-rich brain areas.
- Dopamine antagonists can ameliorate tics.

• Catecholamine depletors (e.g., tetrabenazine) can ameliorate tics.

# 5.2. Background on Ecopipam



Please refer to the Investigator's Brochure for more detailed information about the known benefits and risks of ecopipam.

#### 5.2.2. Clinical Data

#### **5.2.2.1.** Safety in Humans

Clinical Summary: Legacy Schering-Plough Studies in Indications other than TS

The earlier clinical program for ecopipam conducted by Schering-Plough investigated the safety and effectiveness of ecopipam for the treatment of obesity, cocaine addiction, and schizophrenia in adults. These comprised 30 Phase 1 studies; seven Phase 2 pilot studies, 5 in subjects with schizophrenia and 2 (including 1 extension study) in subjects with cocaine addiction; and 1 completed Phase 2 and 3 discontinued Phase 3 studies in subjects with a primary diagnosis of moderate to severe obesity.

The Phase 1 studies examined ecopipam's pharmacokinetics, pharmacodynamics, bioavailability, distribution, food-effects on absorption, interactions with other drugs, bioequivalence of different

formulations, and various physiological effects in cocaine users, smokers, or healthy subjects. The results of these studies demonstrate that ecopipam was well-tolerated with no clinically significant changes in physical examinations, vital signs, electrocardiograms (ECGs), laboratory tests, electroencephalograms (EEGs), neurological examinations, or liver function tests (LFTs). Most of the reported AEs were mild to moderate in intensity. The most commonly reported AE in Phase 1 clinical studies were somnolence. Other commonly reported AEs in Phase 1 clinical studies were headache, fatigue, nausea, and insomnia.

In a Phase 2 study (C197-184), 279 subjects with cocaine dependence in 3 dose groups (10-, 25-, and 100 mg/day) were exposed to ecopipam HCl for 8 weeks in a placebo-controlled study. No differences in the reduction of cocaine use were demonstrated in favor of ecopipam compared with placebo. The most common AEs reported among all subjects in the cocaine addiction studies were fatigue, headache, nausea, insomnia, and somnolence. Fatigue and somnolence appeared to be reported more often in subjects treated with ecopipam than placebo. Somnolence appeared to occur in a dose-related fashion, occurring in 28% (26/94), 31% (29/94), 43% (39/91), and 20% (19/93) of subjects treated with ecopipam HCl 10-, 25-, and 100 mg/day, and placebo, respectively.

Five open-label safety, tolerability and Phase 2 studies of ecopipam in 56 subjects with schizophrenia were conducted. Subjects diagnosed with acute schizophrenia, schizophreniform disorder, or bipolar schizoaffective disorders were treated with ecopipam HCl up to a daily dose of 600 mg. The maximum duration of treatment was 6 weeks. Ecopipam, when administered to subjects with schizophrenia, did not demonstrate efficacy in these studies. The most commonly reported AEs were somnolence (21%, 12/56), headache, nausea, vomiting, and dizziness (each reported in 14%, 8/56 subjects), insomnia (9%, 5/56), dyspepsia (7%, 4/56), and anxiety (7%, 4/56).

In a Phase 2, double-blind, placebo-controlled study (C/I98-271), 185 subjects with a primary diagnosis of moderate to severe obesity were treated with ecopipam HCl (10-, 30-, or 100 mg PO, once per day) for 12 weeks. Subjects receiving ecopipam HCl showed a dose-dependent weight loss. The most commonly reported AEs by subjects receiving ecopipam HCl were headache, 19% (36/185); viral infection, 19% (36/185); somnolence, 18% (34/185); insomnia, 9% (17/185); and nausea, 9% (16/185).

In three Phase 3, double-blind, placebo-controlled studies (P00359, P00396, and P00741), obese subjects including type 2 diabetic subjects were treated with ecopipam HCl (50 or 100 mg PO, once daily [QD]) for 52 weeks. Subjects receiving ecopipam HCl showed a dose-dependent weight loss. These Phase 3 studies were discontinued because of unexpected psychiatric AEs (ecopipam 31% vs. placebo 15%), including depression, anxiety, and suicidal ideation, thereby excluding its projected use in weight management. The most frequently reported AEs in all Phase 3 obesity studies receiving ecopipam HCl were upper respiratory tract infection 30% (439 of 1482 subjects reporting), insomnia 17% (248/1482), headache 16% (244/1482), depression 16% (236/1482), somnolence 15% (216/1482), fatigue 15% (215/1482), anxiety 14% (211/1482), pharyngitis 9% (137/1482), back pain 8% (114/1482), and nausea 7% (107/1482). The frequencies of insomnia, depression, somnolence, and anxiety were about twice as frequent in subjects receiving ecopipam HCl than placebo. The frequencies of upper respiratory tract infection, headache, fatigue, pharyngitis, back pain and nausea were similar in frequencies in subjects receiving ecopipam and placebo.

#### Clinical Summary: Psyadon Studies in Indications other than TS

Following acquisition of ecopipam by Psyadon from Schering-Plough, two Phase 1 studies, one study in Lesch-Nyhan Disease (LND) subjects aged ≥6 years old (PSY101) and one study of the pharmacokinetics of ecopipam controlled release capsules in male adult volunteers (PSY401), were completed.

One Phase 2a study in adult subjects with pathological gambling (PSY201) was also completed. In addition, a Phase 3, multicenter, randomized, double-blind, 3-period crossover study with an open-label extension in subjects with LND ( $\geq$  6 years old) (PSY102) was discontinued before completion for financial (non-safety related) reasons.

In the Phase1 LND study (PSY101), in which 4 of 5 subjects were children, the most commonly reported AEs were sedation (3 subjects), dystonia (2 subjects) and nausea (2 subjects).

In a Phase 2a, single-blind (the subjects were blinded to treatment assignment), nonrandomized study, 28 subjects with pathological gambling (PSY201) received placebo (1-2 tablets/day orally depending on their urge to gamble) for 1 week and then ecopipam HCl (1-2 50-mg tablets/day orally depending on their urge to gamble) for 6 weeks. The most commonly reported AEs (incidence  $\geq$ 5%) were drowsiness (11%), fatigue (11%), anxiety (11%), vomiting (11%), headache (7%), fever (7%), depression (7%), and rhinorrhea (7%).

A Phase 3 study (PSY102) of ecopipam for the treatment of self-injurious behaviors in LND subjects was done. A total of 9 pediatric subjects were enrolled before the study was terminated for non-safety related reasons. Ecopipam HCl was administered at either 50 mg/day (<20 kg body weight) or 100 mg/day (>20 kg body weight). In the PSY102 LND study, 1 subject aged 10 years old experienced dystonia, swallowing difficulty, and depressed mood which involved persistence or significant disability or incapacity. The same subject experienced renal calculus, dystonia, and bronchospasm which involved persistence or significant disability or incapacity, and the relationship to study drug was not related. Another subject aged 6 years old experienced dysphagia, somnolence, and depressed mood which involved persistence or significant disability or incapacity, and the relationship to study drug was possibly related. Since dystonia and dysphagia have not been seen previously in other study populations and because LND subjects have a genetic mutation known to impact dopaminergic systems, it is believed these AEs are uniquely seen in this population and are unlikely to occur in subjects without this disorder.

#### Clinical Summary: Psyadon Clinical Studies in TS Subjects

Two Phase 2 studies in subjects with TS have been conducted.

#### **Study PSY301**

In a Phase 2a multicenter, open-label, nonrandomized study, 18 adult subjects with TS (PSY301) were given ecopipam HCl 50 mg for 2 weeks followed by 100 mg for 6 weeks. The primary outcome measure was Yale Global Tic Severity Score (YGTSS). After ecopipam treatment, YGTSS total score, motor tics score, phonic tics score, and overall impairment were all significantly decreased from baseline to endpoint, which indicated that the severity of tics was decreased. The most commonly reported AEs (incidence 20%) were sedation (33%), insomnia (33%), fatigue (33%), somnolence (28%), headache (22%), muscle twitching (22%), and anxiety (22%).

#### **Study PSY302**

In a Phase 2b multicenter, double blind, randomized, crossover study (PSY302), 40 children/adolescents (ages 7-17 years) were given ecopipam HCl up to 50 mg/day (if <75 lbs) or 100 mg/day (if >75lbs) for 4 weeks. The primary endpoint was the YGTSS Total (MP) Scores which were the sum of the motor and phonic subscales of YGTSS. In the Intent-to-treat (ITT) population, the mean (± standard deviation [SD]) YGTSS Total (MP) Scores at baseline were 32.8 (±7.1) prior to ecopipam treatment and 33.7 (±6.7) prior to placebo treatment. On Day 16 of the treatment period, YGTSS Total (MP) Scores decreased by 5.1 (±8.5) points on ecopipam and 2.1 (±4.7) points on placebo. On Day 30, YGTSS Total (MP) Scores decreased by 5.6 (±8.7) points on ecopipam and 3.4 (±5.8) points on placebo. Similar results were observed in the Evaluable population.

In the ITT population, least square (LS) means (±standard error [SE]) of the difference between ecopipam and placebo treatment were -2.8885±1.5282 (95% confidence interval [CI]: -5.9822, 0.2053, p=0.0664) on Day 16 and -2.1366±1.6551 (95% CI: -5.4871, 1.2139, p=0.2045) on Day 30. The treatment difference was more obvious in the Evaluable population for both days (on Day 16, p=0.0155, and on Day 30, p=0.0435).

With respect to secondary endpoints, the changes of subscale scores were similar to YGTSS Total (MP) Scores results. The secondary endpoints were not ranked in a hierarchical order and multiplicity was not taken into account. In the ITT population, the mean ( $\pm$ SD) motor, phonic, impairment, and global scores (the sum of motor, phonic and impairment scores) at baseline were 18.4 ( $\pm$ 3.3), 14.4 ( $\pm$ 4.9), 28.0 ( $\pm$ 10.7), and 60.8 ( $\pm$ 16.5) prior to ecopipam; and 18.3 ( $\pm$ 3.4), 15.4 ( $\pm$ 4.5), 27.5 ( $\pm$ 9.3), and 61.2 ( $\pm$ 14.0) prior to placebo, respectively. After 30 days of treatment, the decreases in scores compared to baseline were 3.3 ( $\pm$ 4.2), 2.3 ( $\pm$ 4.9), 7.0 ( $\pm$ 11.6), and 12.6 ( $\pm$ 18.7) on ecopipam; and 1.6 ( $\pm$ 3.3), 1.8 ( $\pm$ 3.6), 3.0 ( $\pm$ 9.1), and 6.4 ( $\pm$ 13.4) on placebo, respectively. Similar results were observed in the Evaluable population.

In the ITT population, after 30 days of treatment, Clinician Global Impression (CGI) Severity Scores decreased by  $0.8~(\pm0.7)$  points on ecopipam and  $0.2~(\pm0.9)$  points on placebo. Also, after ecopipam treatment, the percentages of subjects with much improved, minimally improved, no change, minimally worse CGI Improvement ratings were 40.00%, 15.00%, 20.00%, and 12.5%, respectively; while the percentages on placebo were 20.00%, 27.50%, 32.50%, and 12.50%, respectively. Similar results were observed in the Evaluable population. These data suggest that the subjects' disease severity decreased and that they had greater improvement while on ecopipam.

In the ITT population, the mean ( $\pm$ SD) DuPaul ADHD rating scale at baseline was 20.2 ( $\pm$ 11.6) points prior to ecopipam and 22.1 ( $\pm$ 11.3) points prior to placebo. On Day 30, ADHD Scores decreased by 1.9 ( $\pm$ 5.2) points on ecopipam and 2.7 ( $\pm$ 6.6) points on placebo. ADHD scales were almost unchanged after ecopipam treatment. Similar results were observed in the Evaluable population.

In the ITT population, the mean ( $\pm$ SD) YBOCS total scores at baseline were 5.7 ( $\pm$ 6.3) prior to ecopipam and 6.6 ( $\pm$ 6.9) prior to placebo. On Day 30 of the treatment period, YBOCS total scores decreased by 0.8 ( $\pm$ 3.3) points on ecopipam and 0.9 ( $\pm$ 4.1) points on placebo. The results of the obsession and compulsion subscales were similar to the total scores.

The results from the Safety population were the same as the ITT population.

A total of 149 treatment-emergent adverse events (TEAEs) were reported in 35 of the 40 treated subjects (87.50%). There was 1 serious TEAE during placebo treatment and 1 TEAE resulting in dose withdrawn permanently during ecopipam treatment. More patients on placebo had severe adverse events (7.5%) compared to ecopipam (5%). No TEAE resulted in death. There were 20 subjects (50.00%) reporting TEAEs related to study drug during ecopipam treatment and 10 subjects (25.00%) during placebo treatment. Forty percent (40.00%) of TEAEs were mild and 37.50% were moderate. One subject decreased the dosage due to fatigue one day after starting ecopipam. Another subject in the ecopipam group was discontinued from the study due to rash starting at Day 0 of the second treatment phase.

The most common TEAEs during ecopipam treatment were headache (6 of 40), abdominal pain upper (4 of 40), nausea (4 of 40), vomiting (4 of 40), insomnia (4 of 40), and somnolence (4 of 40). The most common TEAEs during placebo treatment were nasopharyngitis (5 of 40), headache (5 of 40), abdominal pain upper (4 of 40), and diarrhea (4 of 40). The most common related TEAEs during ecopipam treatment were nausea (4 of 40) and somnolence (4 of 40). The most common related TEAEs during placebo treatment were headache (3 of 40), somnolence (2 of 40), and initial insomnia (2 of 40).

There was no evidence that administration of ecopipam affected weight, Children's Depression Inventory (CDI) scores or Columbia Suicide Severity Rating Scale (C-SSRS) in the subjects. There were no clinically significant laboratory abnormalities, changes in vital signs, ECG, or physical examination findings after ecopipam administration. There were no AEs related to extrapyramidal reactions.

### 5.3. Risk-Benefit Assessment

A consideration of the potential of risks that TS subjects may be exposed to, approaches to reducing any such risks, and the possible benefits that they may derive from their participation in EBS-101-OL-001 is outlined below.

#### 5.3.1. Assessment of Risk

As 2651 human subjects have been exposed to single and multiple doses ecopipam and safety data including collection of adverse events, physical examinations, laboratory tests, ECGs etc. have been systematically collected, there exists a fair body of information to base the understanding of potential risks and approaches to minimizing them in current and future studies.

Of the 2651 human subjects that have been exposed to ecopipam, 540 adults have participated in studies to investigate the safety, tolerability, pharmacodynamics and pharmacokinetics of ecopipam after single and multiple dose administration. Of the 2651 human subjects that have been exposed to ecopipam, a total of 2058 adult subjects have received treatment with ecopipam in therapeutic studies, including 1667 with obesity, 279 with cocaine addiction, 56 with schizophrenia, schizoaffective disorder and schizophreniform disorder, 28 with pathological gambling, 1 adult with LND, 18 adults with TS, 40 children/adolescents with TS and 9 adults with stuttering. These have shown that ecopipam is generally well tolerated with the adverse events affecting primarily the CNS (e.g., sedation, insomnia, psychiatric changes such as

depression, anxiety and suicidal ideation) and the gastrointestinal system (e.g., nausea and vomiting).

In subjects with TS, ecopipam has been evaluated in two studies, one study in adult subjects with TS and one study in children/adolescents with TS. In the pediatric TS study, overall, adverse events were more common in ecopipam compared to placebo. There were no serious adverse events (SAEs) and only one subject discontinued treatment due to an adverse event in the ecopipam group. Most adverse events were mild to moderate in severity. Adverse events in the Psychiatric Disorders, Central Nervous System Disorders and Gastrointestinal Disorders categories were more common with ecopipam than placebo. Notably, more subjects experienced adverse events of somnolence, insomnia, sedation, restlessness, irritability, nausea and vomiting with ecopipam than with placebo. There were no AEs of extrapyramidal symptoms in the pediatric study. A higher percentage of subjects on ecopipam gained 5 pounds or more during the study than with placebo (17.5% compared to 15%). Orthostatic blood pressure assessments were not done (or not reported). A table of weight changes was provided for the open-label extension study (PSY302A) and almost all of the children gained weight after 3, 6, 9 or 12 months of treatment. Suicidal ideation was seen both during the blinded study as well as the open-label extension study in pediatric subjects on ecopipam. There did not appear to be clinically significant ECG findings. However, open-label extension adverse event data have not yet been analyzed.

In the adult study in TS, the most commonly reported adverse events (incidence  $\geq$ 20%) were sedation (33%), insomnia (33%), fatigue (33%), somnolence (28%), headache (22%), muscle twitching (22%) and anxiety (22%). Two subjects developed adverse event of akathisia and one developed an adverse event of tremor, both of which are extrapyramidal reactions. Three of 18 subjects (16.7%) also discontinued study drug due to an adverse event.

For the older obesity and cocaine dependence program, there were subjects who experienced adverse events of weight gain, suicidal ideation, diabetes, extrapyramidal reactions, somnolence, insomnia, hypotension and sexual side effects. There was no raw data on orthostatic blood pressure. In a table of all adverse events during the whole program, the adverse event of dyskinesia is listed but is not in any of the data tables. When reviewing the large Phase 2 and Phase 3 studies in obesity and the other indications, the rate of tardive dyskinesia appears to be extremely low (or absent) and the rate of other extrapyramidal reactions (akathisia, tremor, etc.) appears at rates that are largely less than what is seen with D1/D2 antagonists. Data for shifts in fasting glucose or lipids were not in the Investigator's Brochure prepared by a previous sponsor and comments were made that there were no significant laboratory changes. There did not appear to be a high rate of increased blood glucose or lipids in the adverse event tables for the other studies. Additionally, data on orthostatic blood pressure changes were not documented but no adverse events of orthostatic hypotension were observed.

#### **5.3.2.** Assessment of Benefit

A review of the efficacy evaluations for ecopipam in the two studies conducted in subjects with TS reveals improvement on the YGTSS scores and other measures of illness severity from baseline to end point.

In a Phase 2a, open-label, non-randomized study (PSY301), the activity and safety of ecopipam in 18 adult subjects with TS was evaluated. Subjects were to receive ecopipam HCl 50 mg for 2 weeks followed by 100 mg for 6 weeks. The primary outcome measure was the YGTSS Total (MP) score. After ecopipam treatment, the YGTSS Total score, motor tics score, phonic tics score and overall impairment decreased from baseline to endpoint, suggesting that the severity of tics was decreased (Table 16, Investigator's Brochure).

In a Phase 2b double-blind, randomized crossover study in children/adolescents (ages 7-17 years) with TS (PSY302), 40 subjects were enrolled and 38 (95.0%) completed the study. The primary endpoint was the YGTSS Total (MP) score.

Ecopipam treatment resulted in a numerical decrease in the YGTSS Total score relative to the placebo treatment, but the decrease was not statistically significant (Figure 9, Investigator's Brochure). The least squares means (±SE) of the difference between ecopipam and placebo treatment were -2.8885 (±1.5282); 95% CI: -5.9822, 0.2053, p=0.0664) on Day 16 and -2.1366 (±1.6551; 95% CI: -5.4871, 1.2139, p=0.2045) on Day 30.

Based on the available safety data, there are some safety advantages for ecopipam compared to D2 antagonists, but the full measure of differentiation will not be known until after a larger and longer Phase 3 program. The rate of tardive dyskinesia and other extrapyramidal reactions commonly associated with D2 antagonists appears much lower with ecopipam. Other possible advantages include a decreased risk of lipid changes, hyperglycemia and orthostatic hypotension.

An individual subject may not receive any therapeutic benefit from participating in an investigational study however, by contributing to medical research, others will be helped. All subjects participating in the study will receive physical examinations, various laboratory tests, ECGs and a systematic evaluation of their condition. Ecopipam may help improve symptoms for participants.

#### **5.3.3.** Methods to Minimize Risks

The following steps are incorporated in the protocol to minimize risks to subjects.

- Subjects will be screened for appropriateness to participate in this study
- All subjects will be evaluated for safety at monthly visits for one year. Follow-up visits will be conducted 7 and 14 days after the last dose of study medication and a follow-up phone call will be conducted 30 days after the last dose of study medication.
- All subjects will be evaluated using the following scales to assess possible worsening of other psychiatric symptoms or other side effects:
  - Abnormal Involuntary Movements Scale
  - Barnes Akathisia Rating Scale
  - Columbia Suicide Severity Rating Scale
  - Children's Depression Rating Scale-Revised
  - Gilles de la Tourette Syndrome Quality of Life Scale

- Pediatric Anxiety Scale
- Clinical Global Impression Tourette Syndrome of Severity

In summary, ecopipam is a new chemical entity with a novel mechanism of action that has some evidence that it may be of therapeutic benefit to subjects with TS. There is also evidence that it is likely to have lower side effect burden (for movement disorders, extrapyramidal symptoms, tardive dyskinesia, etc., metabolic syndrome and elevated prolactin) than the currently used dopamine antagonists. The protocol has processes to minimize potential risks from study medication that participants may be exposed to such that risks from the study balance the potential benefits.

## 6. STUDY OBJECTIVES AND PURPOSE

# 6.1. Primary Objective

The primary objective of this study is to evaluate the long-term safety and tolerability of ecopipam tablets in pediatric subjects (aged  $\geq 6$  to  $\leq 18$  years at Baseline) with TS that were previously enrolled in study EBS-101-CL-001 within the time period specified for this protocol.

# 6.2. Secondary Objectives

The secondary objective of this study is to evaluate the durability of effect of ecopipam in pediatric subjects (aged  $\geq 6$  to  $\leq 18$  years at Baseline) with TS.

### 7. INVESTIGATIONAL PLAN

## 7.1. Overall Study Design

This is an international, multicenter, open-label, long-term extension study evaluating the safety of ecopipam tablets for the treatment of pediatric subjects (aged ≥6 to ≤18 years at Baseline) with TS. Subjects who completed the Phase 2b, randomized, double-blind, efficacy and safety study (EBS-101-CL-001) and who meet all the inclusion/exclusion criteria for this study will be eligible to participate in this study. All subjects will be titrated to a target dose of 2 mg/kg/day as participants rolling over from the Phase 2b double-blind efficacy and safety study will be tapered off of study medication to maintain the blind from that study. Subjects will complete study visits every month for 1 year. A Follow Up visits will be conducted 7 and 14 days after the last dose of study medication and a Follow Up phone call will be conducted 30 days after the last dose of study medication. Study Visits may be completed in locations other than clinic and/or safety and efficacy assessments required at these visits will be made available for remote administration due to restrictions as a consequence of the COVID-19 pandemic or other qualifying event.

Safety will be monitored throughout the study at every visit by repeated adverse event (AE) monitoring, vital signs, the Columbia-Suicide Severity Rating Scale (C-SSRS), the Abnormal Involuntary Movement Scale (AIMS), the Barnes Akathisia Rating Scale (BARS), the Pediatric Anxiety Rating Scale (PARS) and Children's Depression Rating Scale-Revised (CDRS-R). In addition to these assessments, at Baseline, Months 1, 3, 6, 9 and 12 safety will also be monitored by clinical and laboratory evaluations, and electrocardiogram (ECG) monitoring. In addition to the scales aforementioned, the YGTSS, CGI Tourette Syndrome of Severity (CGI-TS-S), and Gilles de la Tourette Syndrome—Quality of Life Scale for Children and Adolescents (C&A-GTS-QOL) will also be assessed at Baseline, Months 1, 3, 6, 9 and 12. The CGI-TS-I will be conducted at Months 1, 3, 6, 9, and 12. At the Follow Up visits, AE monitoring, the C-SSRS, clinical and laboratory evaluations and vital signs will be assessed. A Follow Up phone call will be conducted 30 days after the last dose of study medication to assess AEs.

# 7.2. Number of Subjects

The actual number of subjects that are enrolled will depend on the final number of subjects who complete study EBS-101-CL-001.

# 7.3. Treatment Assignment

Since this is an open-label study, all subjects that have cleared the inclusion/exclusion criteria will be administered ecopipam HCl at a target dose of 2 mg/kg/day.

# 7.4. Dose Adjustment Criteria

Doses will be adjusted based on the following weight bands to better achieve the 2 mg/kg/day target dose:  $\ge 18$  to  $\le 23$  kg, > 23 to  $\le 34$  kg, > 34 to  $\le 44$  kg, > 44 to  $\le 68$  kg, > 68 to  $\le 83$  kg, > 83 kg. Dosing adjustments would be allowed down one dose level based on titration for safety reasons at the discretion of the Principal Investigator. See Section 10.5 for direction on administration of study drug.

# 7.5. Criteria for Subject Study Discontinuation

A subject may elect to discontinue from the study at any time for safety or personal reasons. All subjects who discontinue from the study should complete the early study discontinuation procedures.

Any subject with a new positive response on questions 4 and/or 5 of the C-SSRS will be immediately discontinued and evaluated for risk. Dosing may be restarted at the discretion of the Investigator following consultation with the Sponsor or its designee.

Subjects who discontinue early from the study will be discontinued for one of these primary reasons: AE(s), lost to follow-up, subject choice, inadequate therapeutic effect, and administrative/other. In addition to the primary reason, the subject may have indicated 1 or more of these reasons as secondary reasons for discontinuation. Study disposition information will be collected on the case report form (CRF).

 Table 2:
 Study Design and Schedule of Assessments

| Assessment <sup>4</sup> | Baseline* (Titration) | | | | | Tr | eatmo | End of Study<br>/ Early<br>Termination | Follow Up<br>Visit | Follow Up<br>Phone Call | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Month | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | One and<br>Two Weeks<br>Post Last<br>Dose | 30 Days<br>After Last<br>Dose |
| Study Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 & 15 | |
| Visit Window | | ±3<br>days | ±3 | ±3 | ±3 | ±3<br>days | ±3<br>days | ±3<br>days | ±3<br>days | ±3<br>days | ±3<br>days | ±3<br>days | ±3 <sub>days</sub> | ±3 <sub>days</sub> | ±3days |
| Informed Consent | X | | | | | | | | | | | | | | |
| Inclusion/ Exclusion | X | | | | | | | | | | | | | | |
| Medical/Psychiatric/<br>Medication History | X | | | | | | | | | | | | | | |
| Physical Examination | X | X | | X | | | X | | | X | | | X | X | |
| Vital Signs <sup>1</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| ECG | X | X | | X | | | X | | | X | | | X | | |
| Laboratory Tests<br>(Hematology,<br>Chemistry and<br>Urinalysis) <sup>2</sup> | X | X | | X | | | X | | | X | | | X | X | |
| Urine Drug Screen | X | X | | X | | | X | | | X | | | X | | |
| Urine Pregnancy Test | X | X | | X | | | X | | | X | | | X | | |
| HbA1c | | X | | X | | | X | | | X | | | X | | |
| YGTSS Score | X | X | | X | | | X | | | X | | | X | | |
| CGI-TS-I | | X | | X | | | X | | | X | | | X | | |


| Assessment <sup>4</sup> | Baseline* (Titration) | | | | | Tr | eatm | End of Study<br>/ Early<br>Termination | Follow Up<br>Visit | Follow Up<br>Phone Call | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Month | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | One and<br>Two Weeks<br>Post Last<br>Dose | 30 Days<br>After Last<br>Dose |
| Study Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 & 15 | |
| CGI-TS-S | X | X | | X | | | X | | | X | | | X | | |
| C&A-GTS-QOL | X | X | | X | | | X | | | X | | | X | | |
| Columbia Suicide<br>Severity Rating Scale | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Abnormal Involuntary<br>Movement Scale<br>(AIMS) | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Barnes Akathisia<br>Ratings Scale (BARS) | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Children's Depression<br>Rating Scale-Revised<br>(CDRS-R) | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Pediatric Anxiety<br>Ratings Scale (PARS) | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Adverse Events | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant<br>Medications | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Dispense Study Drug | X | X | X | X | X | X | X | X | X | X | X | X | $X^3$ | | |
| Collect Unused Study<br>Drug/Assess Drug<br>Compliance | | X | X | X | X | X | X | X | X | X | X | X | X | X | |

Confidential

Abbreviations: BP = blood pressure, CGI = Clinician Global Impression, CGI-TS-I = CGI Tourette Syndrome of Improvement, CGI-TS-S = CGI Tourette Syndrome of Severity, ECG = electrocardiogram, HbA1c = Hemoglobin A1c

<sup>\*</sup> Baseline is to occur within 30 days of the EBS-101-CL-001 14 Day Follow Up Visit (or longer with the permission of the medical monitor). All Baseline measurements can be taken from the Day 14 Follow Up Visit of the EBS-101-CL-001 study if performed less than 7 days prior to the Baseline visit. In this case, the HbA1c and Urine Drug Screen from the Week 12/Completion Visit of the EBS-101-CL-001 study may be used.

<sup>&</sup>lt;sup>1</sup> Vital signs will include heart rate, BP, orthostatic BP and heart rate (done supine and then 3 minutes after standing), height and weight.

<sup>&</sup>lt;sup>2</sup> Subjects should be in a fasting state (8 hours) for laboratory tests.

<sup>&</sup>lt;sup>3</sup> Study drug dispensation for down titration.

<sup>&</sup>lt;sup>4</sup> Assessments for Study Visits may be completed in locations other than study clinic and/or safety and efficacy assessments required at these visits will be made available for remote administration due to restrictions as a consequence of the COVID-19 pandemic or other qualifying event.
#### 8. SELECTION AND WITHDRAWAL OF SUBJECTS

## 8.1. Subject Inclusion Criteria

- 1) Subjects must have completed the EBS-101-CL-001 study through the Day 14 Follow Up Visit within the last 30 days (or with permission of the medical monitor) and must be who the Investigator feels would benefit from continued participation.
- 2) Adolescent females of childbearing potential who are sexually active must be using highly effective contraception (i.e., oral contraceptives, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomized male partner) and agree to continue use of highly effective contraception for the duration of their participation in the study. They must also agree to use contraception for 30 days after their last dose of study drug.
- 3) Sexually active male subjects must use a highly effective method of contraception during the study and agree to continue the use of highly effective contraception for at least 30 days after the last dose of study drug.
- 4) Parents or legal guardians of subjects <18 years of age at Baseline must execute a written informed consent. Subjects ≥18 years of age must execute a written informed consent.
- 5) Subjects <18 years of age at Baseline must execute a written informed assent according to the requirements of the site's IRB/EC.

## 8.2. Subject Exclusion Criteria

- 1) Subjects with a clinical presentation and/or history consistent with another neurologic condition that may have had accompanying abnormal movements (e.g., Huntington's disease, Parkinson's disease, Wilson's disease, stroke, Restless Legs Syndrome).
- 2) History of schizophrenia, bipolar disorder, or other psychotic disorders.
- 3) Any unstable primary mood disorder (DSM-5 criteria) at time of Baseline.
- 4) Subjects who have unstable medical illness or clinically significant abnormalities on laboratory tests or ECG at Baseline as determined by the Principal Investigator.
- 5) Subjects who have moderate to severe renal insufficiency at Screening.
- 6) Subjects with a major depressive episode in the past 2 years.
- 7) Subjects with a history of attempted suicide.
- 8) A significant risk of committing suicide based on history, routine psychiatric status examination, Investigator's judgment, or who had an answer of "yes" on any question other than 1–3 (currently or within the past 30 days) on the baseline/screening version of the C-SSRS.
- 9) Subjects with a history of seizures (excluding febrile seizures that occurred <2 years prior to Baseline).
- 10) Subjects with a myocardial infarction within 6 months.

- 11) Female subjects who are currently pregnant or lactating or planning to become pregnant during the course of the study.
- 12) Subjects who have a need for medications which would have unfavorable interactions with ecopipam, e.g., dopamine antagonists or agonists [including bupropion], tetrabenazine, monoamine oxidase inhibitors, or St. John's Wort.
- 13) Subjects with current or recent (past 3 months) DSM-5 substance use disorder (with the exception of nicotine).
- 14) Subjects with positive urine drug screen for cocaine, amphetamine, methamphetamine, benzodiazepines, barbiturates, phencyclidine (PCP) or opiates at Baseline, except those receiving stable, prescribed treatment for ADHD. Subjects with urine positive only for benzodiazepines will be exclusionary unless medically prescribed.
- 15) Subjects with a lifetime history of bipolar disorder type I or II, dementia, schizophrenia, or any other psychotic disorder.
- 16) Inability to swallow tablets.
- 17) Subjects with a known hypersensitivity to ecopipam or any of its excipients.
- 18) Any subject who in the opinion of the investigator is not a suitable candidate for the study.

## 8.3. Subject Withdrawal Criteria

The Investigator or subject themselves may stop study treatment at any time for safety or personal reasons.

Any subject with a CDRS-R assessment indicative of the onset of a new depressive episode at any visit can be discontinued from study participation at the discretion of the Investigator. Any subject with a new positive response on questions 4 and/or 5 of the C-SSRS will be immediately discontinued and evaluated for risk. Dosing may be restarted at the discretion of the Investigator following consultation with the Sponsor or its designee.

Where possible, a subject who discontinues treatment will undergo the protocol-specified end-of study procedures at the time of discontinuation. Date and reason(s) of premature discontinuation will be described on the CRF. In addition, the date of last dose of study treatment will be recorded on the Study Treatment Dosing CRF.

## 9. TREATMENT OF SUBJECTS

## 9.1. Description of Study Drug

**Table 3:** Investigational Product

| | Investigational Product |
|---|---|
| Product Name: | Ecopipam |
| Active Pharmaceutical Ingredient: | Ecopipam hydrochloride |
| Dosage Form: | Tablets |
| Unit Dose (expressed as the free base) | 12.5-, 37.5-, 50-, 75-, and 100 mg |
| Route of Administration | Oral |
| Physical Description | Round, biconvex, light blue film-coated tablet, plain on both sides |
| Manufacturer | Corealis Pharma, Inc. |

#### 9.2. Concomitant Medications

For subjects who receive study treatment, any medication (including over-the-counter medications) administered to the subject during the course of the study (starting at the date of informed consent) will be recorded on the Prior and Concomitant Medication CRF. Nonpharmacologic therapies/procedures will also be captured on the CRF. Non-dopaminergic blocking tic treatment could be allowed in consultation with the PI. The Investigator will record any AE on the Adverse Events CRF for which a concomitant medication was administered.

## 9.3. Prohibited Therapies

Since ecopipam and its metabolite (SCH40853) may inhibit CYP2D6, OATP1B1, PGP and UGT1A9, for any drug that is a substrate of these enzymes, the label for the drug should be consulted to decide if a dose adjustment is needed. Drugs that are strong inducers of these enzymes are prohibited. An illustrative list of such drugs is provided in the Prohibited Medications List in the Appendices.

Prohibited therapies per the exclusion criteria (Section 8.2) include medications which would have unfavorable interactions with ecopipam:

• Dopamine antagonists or agonists (including bupropion)

- Tetrabenazine
- Monoamine oxidase inhibitors
- St. John's Wort

## 9.4. Treatment Compliance

During the study period, subject compliance will be monitored by review of the tablet counts at the study site visits. Any violation of compliance will require evaluation by the Investigator and Sponsor to determine if the subject may continue the study.

## 9.5. Randomization and Blinding

No blinding will be needed as this is an open-label study.

#### 10. STUDY DRUG MATERIALS AND MANAGEMENT

#### 10.1. Study Drug

Ecopipam tablets

## 10.2. Study Drug Packaging and Labeling

Study drug will be supplied in labeled containers by the Sponsor. The product release certificates for ecopipam will be included in the clinical study report for this protocol. Any special storage conditions will be noted on the label and should be followed by the study site.

The labels will be produced by PCI Pharma Services. Minimally, the labels will contain the following information:

- 1. Name, address and telephone number of the Sponsor
- 2. Pharmaceutical dosage form, route of administration, quantity of dosage units, identifier, and dose strength
- 3. Lot number
- 4. Protocol Number
- 5. Study identifier
- 6. Study subject identification number
- 7. Directions of use
- 8. "Caution: New Drug Limited by Federal (US) law to investigational use (or equivalent for rest of world)"
- 9. "Keep out of reach of children"
- 10. Storage Conditions
- 11. Expiration Date

## 10.3. Study Drug Storage

Study drug must be stored as instructed on the study drug label. All relevant site-specific guidelines and country-specific labeling requirements must be followed. Study drug must be kept in a secure location and carefully stored at the study site within its original container and protected from light. A daily temperature log for monitoring of proper storage conditions must be maintained by the site.

## 10.4. Study Drug Preparation

Study drug will be prepared in 15 count bottles for ecopipam.

#### 10.5. Administration

Ecopipam HCl will be supplied as 12.5-, 37,5-, 50-, 75-, and 100-mg tablets. The target dose is 2 mg/kg via oral administration.

During the 4-week titration period, the following ecopipam HCl doses will be administered for each of the weight bands:

- Those who weigh ≥18-≤23 kg will titrate from 12.5 mg daily to 37.5 mg daily: 12.5 mg during Week 1, 25 mg (two 12.5-mg tablets) during Week 2, and 37.5 mg during Weeks 3 and 4.
- Those who weigh >23- $\leq$ 34 kg will titrate from 12.5 mg daily to 50 mg daily: 12.5 mg during Week 1, 25 mg (two 12.5-mg tablets) during Week 2, 37.5 mg during Week 3, and 50 mg during Week 4.
- Those who weigh >34- $\leq$ 44 kg will titrate from 12.5 mg daily to 75 mg daily: 12.5 mg during Week 1, 25 mg (two 12.5-mg tablets) during Week 2, 50 mg during Week 3, and 75 mg during Week 4.
- Those who weigh >44- $\leq$ 68 kg will titrate from 25 mg daily to 100 mg daily: 25 mg (two 12.5-mg tablets) during Week 1, 50 mg during Week 2, 75 mg during Week 3, and 100 mg during Week 4.
- Those who weigh >68- $\leq$ 83 kg will titrate from 25 mg daily to 150 mg daily: 25 mg (two 12.5-mg tablets) during Week 1, 50 mg during Week 2, 100 mg during Week 3, and 150 mg (two 75-mg tablets) during Week 4.
- Those who weigh >83 kg will titrate from 25 mg daily to 200 mg daily: 25 mg (two 12.5-mg tablets) during Week 1, 50 mg during Week 2, 100 mg during Week 3, and 200 mg (two 100-mg tablets) during Week 4.

During the treatment phase, the following ecopipam HCl doses will be administered for each of the weight bands:

- Those who weigh  $\ge 18 \le 23$  kg will receive 37.5 mg daily.
- Those who weigh >23-\(\le 34\) kg will receive 50 mg daily.
- Those who weigh >34-\(\le 44\) kg will receive 75 mg daily.
- Those who weigh >44-\(\le 68\) kg will receive 100 mg daily.
- Those who weigh >68-\le 83 kg will receive 150 mg daily.
- Those who weigh >83 kg will receive 200 mg daily.

All doses will be administered PO once daily in the evening.

At the end of the open-label treatment phase, subjects will titrate off therapy and receive ecopipam HCl doses that will be reduced by 25 mg/day until off of drug; signs of symptoms of withdrawal will be monitored.

Subjects with weight changes during the course of the study resulting in change in weight band may titrate to the dosing of the new weight band at the discretion of the Investigator and with the approval of the Medical Monitor. If approved, the dose of study medication should be increased according to the titration scheme noted for the new weight band.

#### **10.6.** Dosing Rationale

An ecopipam HCl dose of 2 mg/kg/day with titration is targeted in pediatric subjects  $\geq$ 6 to  $\leq$ 18 years of age at Baseline using the dosage regimen proposed in Table 4.

**Table 4:** Proposed Dosing Regimen

| Weight (kg) | Dose (mg)<br>Week 1 | Dose (mg)<br>Week 2 | Dose (mg)<br>Week 3 | Dose (mg)<br>Week 4 onwards |
|---|---|---|---|---|
| ≥18 to ≤23 | 12.5 | 25 (2×12.5) | 37.5 | 37.5 |
| >23 to ≤34 | 12.5 | 25 (2×12.5) | 37.5 | 50 |
| >34 to ≤44 | 12.5 | 25 (2×12.5) | 50 | 75 |
| >44 to ≤68 | 25 (2×12.5) | 50 | 75 | 100 |
| >68 to ≤83 | 25 (2×12.5) | 50 | 100 | 150 (2×75) |
| >83 | 25 (2×12.5) | 50 | 100 | 200 (2×100) |

This dosing regimen was chosen based on modeling and simulation with the results and important information summarized below:

- In a double-blind, placebo-controlled crossover study of 40 subjects with TS aged 7 to 17 years receiving ecopipam HCl at 50 mg (if <75 pounds) or 100 mg (if ≥75 pounds), after a titration, a post-hoc analysis showed that t ecopipam HCl likely has modest efficacy (Study PSY302);
- 2 mg/kg targets a mg/kg dose that is above the median mg/kg dose in 75% of subjects in Study PSY302, with the remaining 25% of subjects having a mg/kg dose that is substantially below the 95<sup>th</sup> percentile from Study PSY302;
- The predicted plasma concentration-time curves for the median, 5<sup>th</sup> percentile, and 95<sup>th</sup> percentile are within the exposures studied in PSY302, and similar to other proposed dosing regimens;
- The animal:human ratios for the active moieties (unconjugated parent plus active metabolite, SCH40853) are adequate based on the no-observed-adverse-effects-level (NOAEL) in the 3-month GLP toxicology study for mice (30 mg/kg), the 3-month GLP toxicology study in rhesus monkeys at 12 mg/kg, and the 1-year GLP toxicology study in cynomolgus monkeys at 12 mg/kg, and do not differ from those in Study PSY302 (Table 5).
- For rhesus and cynomolgus monkeys, the main toxicities observed at 12 mg/kg were decreased activity, decreased appetite, and decreased defecation. For cynomolgus monkeys, these AEs were reported during the first 1 to 3 weeks (hence, the need for titration in the proposed clinical study Protocol EBS-101-OL-001).
- In Study PSY302, the TEAEs were gastrointestinal disorders (e.g., nausea, upper abdominal pain), general disorders and administrative site conditions (e.g., decreased appetite, fatigue), and nervous systems disorders (e.g., somnolence, headache, sedation). The current study will incorporate a 2-week titration which has the potential to improve tolerability.

• While studying multiple dose levels is important in a Phase 2b study, a dose titration approach (instead of fixed 3-dose parallel design study) was chosen because the PSY302 study suggested that doses lower than ~1.4 mg/kg the 25<sup>th</sup> percentile would be unlikely to have substantial efficacy. The exposure between ~1.4 mg/kg and ~2 mg/kg would have significant overlap in exposure (i.e., they would not be distinctly different doses), doses higher than ~2 mg/kg may not be well tolerated, and doses higher than ~2 mg/kg would result in animal:human exposures significantly lower than 1.

Table 5: Animal:Human Exposure Ratios with the Proposed Dosage Regimen of Ecopipam HCl to 7 to 16 Year Olds

| Week | PK | Mice:<br>Human<br>Ratio <sup>b,c</sup> | Rhesus Monkey:<br>Human Ratio <sup>c</sup> | | Cynomolgus<br>Human | • |
|---|---|---|---|---|---|---|
| | | 30 mg/kg | 3 mg/kg | 12 mg/kg | 3 mg/kg | 12 mg/kg |
| Combine | ed AUC <sup>a</sup> (1 | ng*hr/mL) | | | | |
| 1 | 146 | 17.2× | 2.1× | 5.9× | 2.1× | 10.6× |
| 2 | 289 | 8.7× | 1.1× | 3.0× | 1.1× | 5.3× |
| Full<br>Dose | 535 | 4.7× | 0.6× | 1.6× | 0.6× | 2.9× |
| Combine | ed C <sub>max</sub> a (n | ig/mL) | | | | |
| 1 | 17.1 | 16.9× | 1.4× | 3.4× | 1.5× | 8.7× |
| 2 | 34.3 | 8.4× | 0.7× | 1.7× | 0.8× | 4.3× |
| Full<br>Dose | 62.6 | 4.6×° | 0.4× | 0.92× | 0.4× | 2.4×° |

 $<sup>^{\</sup>rm a}$  Animal: human ratios were calculated based on combined unconjugated parent ecopipam HCl plus active metabolite SCH40853 AUC and  $C_{\rm max}$ .

 $<sup>^</sup>b$  The ratios for rats at 6 mg/kg are not included due to the fact that the assay sensitivity was not adequate (LLOQ=0.5 μg/mL), the AUC was determined with ≤3 data points, and there were too few concentrations above the LLOQ to determine the  $C_{max}$ 

<sup>&</sup>lt;sup>c</sup> Ratios were calculated using the predicted exposure in Study PSY302. These animal:human ratios did not differ in most cases for the full dose where the animal:human C<sub>max</sub> ratios differed by 0.1 times where noted.

#### 10.7. Study Drug Accountability

The Investigator (or pharmacist, as appropriate) must maintain records of the delivery of the study drug to the study site, the inventory at the site, use for each subject, and return of the study drug to a delegate of the Sponsor. Total study site accountability will be conducted at the end of the study and the Investigator must explain all discrepancies.

A Drug Dispensing Log must be kept current and should contain the following information:

- Identification (subject number and initials as required by local regulations) of subject to whom the study drug was dispensed
- The dates and lot numbers for the study drug dispensed
- Initial inventory on receipt of drug at the site
- Final inventory on completion of the study

All records and inventory must be available for inspection by the Clinical Research Associate (CRA).

Due to the COVID-19 pandemic, in some cases direct to patient shipments may be necessary. In this case, study medication may be transported to the subject by a third party vendor who has systems in place to protect patient privacy and data integrity. On close-out of the site, all used and unused investigational product must be shipped to the Emalex-designated location. The Drug Dispensing Log must be available for monitoring, auditing, or inspection.

## 10.8. Study Drug Handling and Disposal

Current ICH Good Clinical Practices (GCP) Guidelines require the Investigator to ensure that study drug deliveries from the Sponsor are received by a responsible person (e.g., pharmacist), and

- That such deliveries are recorded
- That study drug is handled and stored safely and properly
- That study drug is only dispensed to study subjects in accordance with the protocol
- That any unused study drug is returned to the Sponsor or standard procedures for the alternative disposition of unused study drug are followed.

#### 11. ASSESSMENT OF EFFICACY

Assessments may be completed in locations other than study clinic and/or via remote administration due to restrictions as a consequence of the COVID-19 pandemic or other qualifying event.

#### 11.1 Efficacy Assessments

The YGTSS, CGI-TS-S, and C&A-GTS-QOL will be assessed at Baseline, Months 1, 3, 6, 9 and 12. The CGI-TS-I will be assessed at Months 1, 3, 6, 9 and 12.

The YGTSS is a clinician-completed rating scale used to quantify overall tic severity as well as specific subdomains of tic number, frequency, duration, intensity, and complexity. Each of these subdomains is scored, on a 5-point scale, separately for motor and vocal tics and then summed across both motor and vocal tics to yield a tic severity score ranging from 0 to 50. The YGTSS also provides for an overall impairment rating (0 = "none" to 50 = "severe"). The YGTSS has demonstrated acceptable internal consistency, good interrater reliability, and acceptable convergent and divergent validity. Efficacy will be analyzed for both the YGTSS-TTS and Global YGTSS.

The CGI consists of 2 reliable and valid 7-item Likert scales used to assess severity and change in clinical symptoms. The scale ranges from 1 = "very much improved" to 7 = very much worse" for the CGI-TS-I. The CGI severity scale (CGI-TS-S) will be used at each study site visit and ranges from 1 = "not ill at all" to 7 = "among the most extremely ill."

Gilles de la Tourette Syndrome—Quality of Life Scale for Children and Adolescents (C&A-GTS-QOL) is a patient-reported health related quality of life measure developed for children and adolescents. Versions of the scale appropriate for subjects 6-12 years of age and 13-18 years of age will be provided. Subjects who turn 13 during the course of the study should continue to be assessed using the version of the scale initially administered.

#### 12. ASSESSMENT OF SAFETY

#### 12.1. Safety Parameters

Study Visits may be completed in locations other than clinic and/or via remote administration due to restrictions as a consequence of the COVID-19 pandemic or other qualifying event. Safety will be monitored throughout the study at all visits by repeated adverse event (AE) monitoring, vital signs, the Columbia-Suicide Severity Rating Scale (C-SSRS), the Abnormal Involuntary Movement Scale (AIMS), the Barnes Akathisia Rating Scale (BARS), the Pediatric Anxiety Rating Scale (PARS) and Children's Depression Rating Scale-Revised (CDRS-R). In addition to these assessments, at Baseline, Months 1, 3, 6, 9 and 12 safety will also be monitored by clinical and laboratory evaluations and electrocardiogram (ECG) monitoring. At the Follow Up visit, AE monitoring, the C-SSRS, clinical and laboratory evaluations and vital signs will be assessed. Laboratory evaluations will include hematology, chemistry, urine values and HbA1c. A Follow Up phone call will be conducted 30 days after the last dose of study medication to assess AEs. Additional assessments (all visits except the follow up visit) will include the AIMS, the BARS, the CDRS-R and the PARS. C-SSRS will also be assessed (all visits including the Follow Up visit).

The C-SSRS is a low burden (approximately 5 minutes for completion) instrument to assess both suicidal behavior and ideation. The scale is appropriate for subjects from age 6 through to an elderly population.

The AIMS records the occurrences of tardive dyskinesia (TD) in subjects receiving neuroleptic medications. The test is used to detect TD and to follow the severity over time.

Barnes Akathisia Rating Scale (BARS) scale to assess the severity of drug-induced akathisia. Objective and subjective items in the scale measure the level of subject's restlessness.

Children's Depression Rating Scale-Revised (CDRS-R) is a clinically validated rating scale designed to assess psychiatric signs and symptoms of depressions in children and adolescents.

Pediatric Anxiety Rating Scale (PARS) is a clinician-rated instrument for assessing the severity of anxiety symptoms associated with common anxiety disorders and generalized anxiety in children and adolescents.

#### **Vital Signs:**

Vital signs will be collected each clinic visit. They include heart rate, blood pressure, orthostatic blood pressure and heart rate (after being supine for 5 minutes and 3 minutes after standing), height and weight.

#### **Clinical Laboratory Assessments:**

The following clinical laboratory tests will be performed in a fasting state at Baseline, Months 1, 3, 6, 9 and 12:

#### **Clinical Laboratory Tests**

<u>Category</u> <u>Parameters</u>

Hematology Red blood cell count, hemoglobin,

hematocrit, platelets, and white blood cell count with differential (neutrophils, bands lymphocytes, monocytes, eosinophils,

basophils)

Chemistry

Electrolytes Sodium, potassium, chloride, bicarbonate

Liver function tests

Alkaline phosphatase, aspartate

aminotransferase (AST), alanine

aminotransferase (ALT), total bilirubin,

direct bilirubin

Renal function parameters Blood urea/blood urea nitrogen (BUN),

creatinine

Other Glucose, calcium, albumin, cholesterol,

triglycerides, phosphorus, lactate dehydrogenase (LDH), total protein,

globulin

Urinalysis Complete urinalysis includes color,

appearance, specific gravity, pH, protein,

glucose, ketones, and blood with microscopic examination for positive

protein or blood results

Pregnancy Test Urine test (for women of childbearing

potential only)

**Special Parameters - Hemoglobin** 

A1c (HbA1c)

#### **Contraception Guidelines:**

As specified in the Inclusion Criteria (Section 8.1), adolescent females of childbearing potential who are sexually active and male subjects who are sexually active must use a highly effective form of contraception throughout the study and for 30 days after the last dose of study drug. See the Contraception Guidelines for additional information.

Subjects must be monitored for signs of study drug abuse, and withdrawal or dependence and if detected must be recorded as AEs.

#### 12.2. Adverse and Serious Adverse Events

#### 12.2.1. Definition of Adverse Events

An AE is defined as any untoward medical occurrence in a subject administered a study drug and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not related to the study

drug. In clinical studies, an AE can include an undesirable medical condition occurring at any time, including baseline or washout periods, even if no study treatment has been administered.

An abnormality identified during a medical test (e.g., laboratory parameter, vital sign, ECG data, physical examination) should be defined as an AE only if the abnormality meets one of the following criteria:

- Induces clinical signs or symptoms
- Requires active intervention
- Requires interruption or discontinuation of study medication
- The abnormality or investigational value is clinically significant in the opinion of the Investigator

All AEs that occur after any subject has been screened, enrolled, before treatment, during treatment, or within 30 days following the cessation of treatment, whether or not they are related to the study, must be recorded on forms provided by the Sponsor or its representative.

#### 12.2.1.1. Treatment-Emergent Adverse Event

A TEAE is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered casually related to the product.

#### 12.2.1.2. Serious Adverse Event

An SAE is an AE occurring during any study phase (i.e., baseline, treatment, washout, or followup), and at any dose of the investigational product, comparator or placebo, that fulfils one or more of the following:

- It results in death
- It is immediately life-threatening
- It requires in-patient hospitalization or prolongation of existing hospitalization
- It results in persistent or significant disability or incapacity
- It results in a congenital abnormality or birth defect
- It is an important medical event that may jeopardize the subject or may require medical intervention to prevent one of the outcomes listed above.

All SAEs that occur after any subject has been enrolled, before treatment, during treatment, or within 30 days following the cessation of treatment, whether or not they are related to the study, must be recorded on forms provided by the Sponsor or its representative.

#### 12.2.1.3. Other Adverse Event

Other AEs (OAEs) will be identified by the Drug Safety Physician and if applicable, also by the Clinical Study Team Physician, during the evaluation of safety data for the clinical study report. Significant AEs of particular clinical importance, other than SAEs and those AEs leading to discontinuation of the subject from the study, will be classified as OAEs. For each OAE, a

narrative may be written and included in the clinical study report. Adverse events of special interest (AESI) are listed in Section 13.2.1.

## 12.3. Relationship to Study Drug

An Investigator who is qualified in medicine must make the determination of relationship to the investigational product for each AE (Unrelated, Possibly Related, or Probably Related). The Investigator should decide whether, in his or her medical judgment, there is a reasonable possibility that the event may have been caused by the investigational product. If no valid reason exists for suggesting a relationship, then the AE should be classified as "Unrelated." If there is any valid reason, even if undetermined, for suspecting a possible cause-and-effect relationship between the investigational product and the occurrence of the AE, then the AE should be considered "Related."

If the relationship between the AE/SAE and the investigational product is determined to be "possible" or "probable", the event will be considered to be related to the investigational product for the purposes of expedited regulatory reporting.

### 12.4. Recording Adverse Events

Adverse events spontaneously reported by the subject and/or in response to an open question from the study personnel or revealed by observation will be recorded during the study at the investigational site. Clinically significant changes in laboratory values, blood pressure, and pulse rate need not be reported as AEs per the Investigator's judgement. However, abnormal values that constitute an SAE or lead to discontinuation of administration of study drug must be reported and recorded as an AE. Information about AEs and SAEs will be collected from the signing of the informed consent form until 30 days following the last dose of study drug. The S/AE term should be reported in standard medical terminology when possible. For each S/AE, the Investigator will evaluate and report the onset (date and time), resolution (date and time), intensity, causality, action taken, serious outcome (if applicable), and whether or not it caused the subject to discontinue the study/study treatment.

Intensity will be assessed according to the following scale:

- Mild (awareness of sign or symptom, but easily tolerated)
- Moderate (discomfort sufficient to cause interference with normal activities)
- Severe (incapacitating, with inability to perform normal activities)

It is important to distinguish between serious and severe AEs. Severity is a measure of intensity, whereas seriousness is defined by the criteria under Section 12.2.1.2. An AE of severe intensity may not be considered serious.

Should a pregnancy of a subject or partner occur, it must be reported and recorded on the Sponsor or its representatives' pregnancy form. Pregnancy in itself is not regarded as an AE unless there is a suspicion that the investigational product may have interfered with the effectiveness of a contraceptive medication. Reports of pregnancy must be submitted to Syneos Health Safety & Pharmacovigilance within one business day:

Email Address: SafetyPV@syneoshealth.com

Fax no. Americas: +1 866 856 1649

Fax no. Europe and ROW +44 1628 461184

The outcome of all pregnancies (spontaneous miscarriage, elective termination, normal birth or congenital abnormality) must be followed up and documented even if the subject was discontinued from the study.

All reports of congenital abnormalities/birth defects are SAEs. Spontaneous miscarriages should also be reported and handled as SAEs. Elective abortions without complications should not be handled as AEs.

## 12.5. Reporting Adverse Events

All SAEs (related and unrelated) will be recorded from the signing of consent form until 30 days following the end of treatment exposure. Any SAEs considered possibly or probably related to the investigational product and discovered by the Investigator at any time after the study should be reported. All SAEs must be reported to Syneos Health Safety & Pharmacovigilance within 1 business day of the first awareness of the event:

Email Address: SafetyPV@syneoshealth.com

Fax no. Americas: +1 866 856 1649

Fax no. Europe and ROW +44 1628 461184

The Investigator must complete, sign and date the SAE pages, verify the accuracy of the information recorded on the SAE pages with the corresponding source documents, and send a copy to the Sponsor or its representatives. Additional follow-up information, if required or available, should all be sent to the Sponsor or its representatives within 1 business day of receipt, and this should be completed on a follow-up SAE form and placed with the original SAE information and kept with the appropriate section of the CRF and/or study file.

The Sponsor and its representatives are responsible for notifying the relevant regulatory authorities of certain events. It is the Principal Investigator's responsibility to notify the Institutional Review Board (IRB) or Independent Ethics Committee (IEC) of all SAEs that occur at his or her site. Investigators will also be notified of all unexpected and serious, drug-related events (7/15 Day Safety Reports) that occur during the clinical study. Each site is responsible for notifying its IRB or IEC of these additional SAEs.

#### 13. STATISTICS

All data analyses will be performed by the Sponsor or its representatives after the study is completed and the database is finalized and released. The statistical analyses described in this section will be performed using SAS 9.4 or higher. Additional analyses may need to be conducted for data not collected at sites and/or via remote administration due to restrictions as a consequence of the COVID-19 pandemic or other qualifying event, these additional analyses will be specified in the SAP.

## 13.1. Analysis Populations

The Safety Population will include all subjects who received at least one dose of study drug from the open labeled study. The Safety Population will be used for the analysis of the safety endpoints.

The Intent-to-Treat (mITT) Population will consist of all subjects who receive at least one dose of study drug. All efficacy analyses will be conducted using the mITT population.

## 13.2. Planned Analyses

#### 13.2.1. Safety Analysis

Adverse Events:

AEs, which include clinical laboratory test variables, will be documented from the time of the first study medication administration from the open label study until the subject's study participation is complete (study discontinuation and up to 30-days follow-up). All AEs that occur after the first study medication application and up to 30 days after the subject's last study medication application will be considered TEAEs.

Each AE will be reported with severity (mild, moderate, severe), seriousness, duration, resolution, action taken, and its relationship with the study medication (related or not related).

Adverse events will be summarized using system organ classification (SOC) defined by Medical Dictionary for Regulatory Activities (MedDRA); the following AEs will be categorized as AESIs in this study (AEs fitting under these categories to be fully described in the SAP):

- Extrapyramidal reactions (i.e. tardive dyskinesia, akathisia)
- Metabolic changes (hyperglycemia/diabetes mellitus, dyslipidemia, weight gain)
- Orthostatic hypotension
- Suicidality
- Leukopenia, neutropenia, agranulocytosis

TEAEs and AESIs will be summarized by severity and by relationship to study medication. Serious TEAEs and TEAEs leading to study termination will be summarized separately.

Other Safety Assessments:

Laboratory values, vital signs, ECG, and physical examination will be summarized descriptively by visit.

#### 13.2.2. Efficacy Analysis

The efficacy outcome measures will be measured at Baseline, Months, 1, 3, 6, 9, and 12 which is end of study or early termination; and include:

- YGTSS-TTS, which is the combined score from the motor and phonic tic score,
- YGTSS Impairment score and global YGTSS (YGTSS-TTS + Impairment score),
- CGI-TS-S
- CGI-TS-I (not measured at Baseline)

The observed YGTSS-TTS, YGTSS-Global and CGI values and their changes from baseline will be summarized by visit. The paired t-test may be used for analyzing the change from baseline within treatment.

The CGI-TS-S, CGI-TS-I and C&A-GTS-QOL values will also be summarized descriptively by visit as continuous and categorical variables.

#### 14. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

## 14.1. Study Monitoring

Before an investigational site can enter a subject into the study, a representative of the Sponsor will visit the investigational study site to:

- Determine the adequacy of the facilities
- Discuss with the Investigator(s) and other personnel their responsibilities with regard to protocol adherence, and the responsibilities of Emalex or its representatives. This will be documented in a Clinical Study Agreement between Emalex and the Investigator.

During the study, a monitor from Emalex or its representative will have regular contacts with the investigational site, for the following:

- Provide information and support to the Investigator(s)
- Confirm that facilities remain acceptable
- Confirm that the investigational team is adhering to the protocol, that data are being accurately recorded in the case report forms, and that investigational product accountability checks are being performed
- Perform source data verification. This includes a comparison of the data in the CRFs with the subject's medical records at the hospital or practice, and other records relevant to the study. This will require direct access to all original records for each subject (e.g., clinic charts).
- Record and report any protocol deviations not previously sent to Emalex.
- Confirm AEs and SAEs have been properly documented on the applicable CRFs and confirm any SAEs have been forwarded to Emalex and those SAEs that met criteria for reporting have been forwarded to the IRB.

The monitor will be available between visits if the Investigator(s) or other staff needs information or advice.

## 14.2. Audits and Inspections

Authorized representatives of Emalex, a regulatory authority, or an IEC/IRB may visit the site to perform audits or inspections, including source data verification. The purpose of an Emalex audit or inspection is to systematically and independently examine all study-related activities and documents to determine whether these activities were conducted, and data were recorded, analyzed, and accurately reported according to the protocol, ICH GCP, and any applicable regulatory requirements. The Investigator should contact Emalex immediately if contacted by a regulatory agency about an inspection.

# 14.3. Institutional Review Board (IRB)/Independent Ethics Committee (IEC)

IRB/IEC approval for the investigation must be obtained prior to initial dosing of any subjects. Initial IRB/IEC approval, and all materials approved by the IRB/IEC for this study, including the subject informed consent form and recruitment materials, must be maintained by the Investigator and made available for inspection.

The Investigator shall make accurate and adequate written progress reports to the IRB/IEC at appropriate intervals, not exceeding 1 year. The Investigator shall make an accurate and adequate final report to the IRB/IEC within 90 days after the close-out visit or within 1 year after last patient out (LPO) or termination of the study, whichever is earlier.

## 15. QUALITY CONTROL AND QUALITY ASSURANCE

To ensure compliance with GCP and all applicable regulatory requirements, Emalex or its designee may conduct a quality assurance audit. Please see Section 14.2 for more details regarding the audit process.

The Sponsor implements and maintains quality assurance and quality control systems in accordance with written SOPs to ensure that studies are conducted and data are generated, documented (record), and reported in compliance with the protocol, GCP, and applicable regulatory requirement(s).

The Sponsor or its representative may arrange to inspect/audit the clinical study at any or all investigational sites. The auditor is independent from the Sponsor's clinical monitoring and project management team. The audit may include on-site review of regulatory documents, CRFs, and source documents. Direct access to these documents will be required by the auditors.

#### 16. ETHICS

#### 16.1. Ethics Review

The final study protocol, including the final version of the informed consent form, must be approved or given a favorable opinion in writing by an IRB or IEC, as appropriate. The Investigator must submit written approval to Emalex before he or she can enroll any subject into the study.

The Principal Investigator is responsible for informing the IRB or IEC of any amendment(s) to the protocol in accordance with local requirements. In addition, the IRB or IEC must approve all advertising used to recruit subjects for the study. The protocol must be re-approved by the IRB or IEC upon receipt of amendments and annually, as local regulations require.

The Principal Investigator is also responsible for providing the IRB with reports of any reportable serious adverse drug reactions from any other study conducted with the investigational product. Sponsor or its representative will provide this information to the Principal Investigator.

Progress reports and notifications of serious adverse drug reactions will be provided to the IRB or IEC according to local regulations and guidelines.

## 16.2. Ethical Conduct of the Study

The study will be performed in accordance with ethical principles that have their origin in the Declaration of Helsinki and are consistent with ICHGCP, applicable regulatory requirements, and Sponsor's policy on Bioethics.

#### 16.3. Written Informed Consent

The Principal Investigator(s) at each center will ensure that the subject and his/her parents or legal guardian is given full and adequate oral and written information about the nature, purpose, possible risk and benefit of the study. Subjects and their parents or legal guardian must also be notified that subjects are free to discontinue from the study at any time. The subject and his/her parents or legal guardian should be given the opportunity to ask questions and allowed time to consider the information provided.

For subjects <18 years of age at Baseline, the parents' or legal guardian's signed and dated informed consent and the subject's signed and dated assent form must be obtained before conducting any study procedures. Subject assents will be administered according to the requirements of the site's IRB/EC. Subjects ≥18 years of age must execute a written informed consent.

The Principal Investigator(s) must maintain the original, signed informed consent form and assent form. A copy of the signed informed consent form and assent form must be given to the subject and his/her parents or legal guardian.

## 16.4. Subject Confidentiality

The information obtained during the conduct of this clinical study is confidential, and disclosure to third parties, other than those noted below, is strictly prohibited. Upon the subject's and

his/her parents' or legal guardian's permission, medical information may be given to his or her personal physician or other appropriate medical personnel responsible for his or her medical welfare.

The Sponsor will use the information obtained during the conduct of this trial for the development of ecopipam. The study Investigator is obliged to provide the Sponsor with complete test results and all data developed in this study, as described in this protocol.

Monitors, auditors, and other authorized agents of the Sponsor and/or its designee, the IEC(s)/IRB(s) approving this research, and competent authority in each participating country, as well as that of any other applicable agency(ies), will be granted direct access to the subjects' original medical records for verification of clinical study procedures and/or data, without violating the confidentiality of the subjects, to the extent permitted by the law and regulations. In any presentations of the results of this study or in publications, the subjects' identity will remain confidential.

#### 17. DATA HANDLING AND RECORDKEEPING

## 17.1. Inspection of Records

Sponsor or its representative will be allowed to conduct site visits at the investigation facilities for the purpose of monitoring any aspect of the study. The Investigator agrees to allow the monitor to inspect the drug storage area, study drug stocks, drug accountability records, subject charts and study source documents, and other records relative to study conduct.

#### 17.2. Retention of Records

The Principal Investigator must maintain all documentation relating to the study for a period of 2 years after the last marketing application approval, or if not approved, 2 years following the discontinuation of the test article for investigation. If it becomes necessary for Emalex or the regulatory authority to review any documentation relating to the study, the Investigator must permit access to such records.

#### 18. PUBLICATION POLICY

The treating physician is obliged to provide the Sponsor with complete data derived from the program. During the program, only Emalex Biosciences may make information available to other participating physicians or to regulatory agencies, except as required by law or regulation. Except as otherwise allowable in the Clinical Site Agreement, any public disclosure (including publicly accessible websites) related to the protocol or program results, is the sole responsibility of Emalex Biosciences.

Emalex Biosciences may publish any data and information from the program (including data and information generated by the physicians) without the consent of the treating physician. Manuscript authorship for any peer-reviewed publication will appropriately reflect contributions to the production and review of the document. All publications and presentations must be prepared in accordance with this section and the Clinical Site Agreement. In the event of any discrepancy between the protocol and the Clinical Site Agreement, the Clinical Site Agreement will prevail. All scientific publications generated by Emalex Biosciences and its agents will be consistent with the principles outlined in Good Publication Practices.

Data from all sites participating in the program will be pooled and analyzed by Emalex Biosciences or its representatives. The first publication of the results shall be made in conjunction with the results from other sites as a multicenter publication. If a multicenter publication is not forthcoming within 24 months of completion of the program at all sites, the treating physician may publish or present the results generated at his or her site.

The treating physician will provide Emalex Biosciences with a copy of any proposed publication or presentation for review and comment at least 60 days prior to such presentation or submission for publication. Emalex Biosciences shall inform the Investigator in writing of any changes or deletions in such presentation or publication required to protect Emalex Biosciences' confidential and proprietary technical information and to address inaccurate data or inappropriate interpretations in the context of any pooled multicenter results. At the expiration of such 60-day period, the physician may proceed with the presentation or submission for publication unless Emalex Biosciences has notified the institution or the physician in writing that such proposed publication or presentation discloses Emalex Biosciences' confidential and proprietary technical information. Further, upon the request of Emalex Biosciences, the physician will delay the publication or presentation for an additional 90 days to permit Emalex Biosciences to take necessary actions to protect its intellectual property interests.

#### 19. LIST OF REFERENCES

- 1. Leckman JF, Bloch MH, Scahill L, and King RA. Tourette syndrome: The self under siege. J Child Neurol 2006;21:642-649.
- 2. Gaze C, Kepley HO, and Walkup JT. Co-occurring psychiatric disorders in children and adolescents with Tourette's syndrome. J Child Neurol 2006;21:657-664.
- 3. Leckman JF. Phenomenology of tics and natural history of tic disorders. Brain Devel 2003;25(S1):S24-S28.
- 4. Keen-Kim D and Freimer NB. Genetics and epidemiology of Tourette syndrome. J Child Neurol 2006;21:665-671.
- 5. Srour M, Lesperance P, Richer F, and Chouinard S. Pediatric psychopharmacology: psychopharmacology of tic disorders. J Can Aca Child Adolesc Psychiatry 2008;17:150-159.
- 6. Harris K and Singer HS. Tic disorders: Neural circuits, neurochemistry, and neuroimmunology. J Child Neurol 2006;21:678-689.
- 7. Mink JW. Basal ganglia dysfunction in Tourette's syndrome: A new hypothesis. Pediatr Neurol 2001;25:190-198.

## 20. REFERENCES FOR QUESTIONNAIRES AND SCALES

- 1. Leckman JF, Riddle MA, Hardin MT, Ort SI, Swartz KL, Stevenson J, et al. The Yale Global Tic Severity Scale: initial testing of a clinician-rated scale of tic severity. J Am Acad Child Adolesc Psychiatry 1989;28(4):566-73
- 2. Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77
- 3. Leckman JF, Towbin KE, Ort SI, Cohen DJ. Clinical assessment of tic disorders severity. In: Cohen DJ, Bruun RD, Leckman JF, editors. Tourette's Syndrome and Tic Disorders: Clinical Understanding and Treatment. New York: John Wiley & Sons; 1988
- 4. Guy, William (1976). "Clinical Global Impressions". ECDEU Assessment Manual for Psychopharmacology—Revised. Rockville, MD: U.S. Department of Health, Education, and Welfare; Public Health Service, Alcohol; Drug Abuse, and Mental Health Administration; National Institute of Mental Health; Psychopharmacology Research Branch; Division of Extramural Research Programs
- 5. Abnormal involuntary movement scale [AIMS] (1976). National Institute of Mental Health Psychopharmacology Research Branch. Guy, W. (1976). ECDEU assessment manual for psychopharmacology. Rev. Rockville, MD: U.S. National Institute of Health, Psychopharmacology Research Branch. Pg. 534-537
- 6. Barnes T.R. A rating scale for drug-induced akathisia. British Journal of Psychiatry. 1989;154:672-676.
- 7. Poznanski EO, Freeman LN, Mokros HB. Children's Depression Rating Scale Revised (September 1984). Psychopharmacol Bull 1985; 21:979-989.
- 8. Su M, McFarlane F, Cavanna A, et al. The English Version of the Gilles de la Tourette Syndrome–Quality of Life Scale for Children and Adolescents (C&A-GTS-QOL). J Child Neurol 2017;32(1):76-83.
- 9. Research Units on Pediatric Psychopharmacology Anxiety Study Group. The Pediatric Anxiety Rating Scale (PARS): development and psychometric properties. J Am Acad Child Adolesc Psychiatry 2002;41;1061-9.

#### 21. APPENDICES

## WMA DECLARATION OF HELSINKI – ETHICAL PRINCIPLES FOR MEDICAL RESEARCH INVOLVING HUMAN SUBJECTS

#### **Preamble**

1. The World Medical Association (WMA) has developed the Declaration of Helsinki as a statement of ethical principles for medical research involving human subjects, including research on identifiable human material and data.

The Declaration is intended to be read as a whole and each of its constituent paragraphs should be applied with consideration of all other relevant paragraphs.

2. Consistent with the mandate of the WMA, the Declaration is addressed primarily to physicians. The WMA encourages others who are involved in medical research involving human subjects to adopt these principles.

## **General Principles**

- 3. The Declaration of Geneva of the WMA binds the physician with the words, "The health of my patient will be my first consideration," and the International Code of Medical Ethics declares that, "A physician shall act in the patient's best interest when providing medical care."
- 4. It is the duty of the physician to promote and safeguard the health, well-being and rights of patients, including those who are involved in medical research. The physician's knowledge and conscience are dedicated to the fulfilment of this duty.
- 5. Medical progress is based on research that ultimately must include studies involving human subjects.
- 6. The primary purpose of medical research involving human subjects is to understand the causes, development and effects of diseases and improve preventive, diagnostic and therapeutic interventions (methods, procedures and treatments). Even the best proven interventions must be evaluated continually through research for their safety, effectiveness, efficiency, accessibility and quality.
- 7. Medical research is subject to ethical standards that promote and ensure respect for all human subjects and protect their health and rights.
- 8. While the primary purpose of medical research is to generate new knowledge, this goal can never take precedence over the rights and interests of individual research subjects.
- 9. It is the duty of physicians who are involved in medical research to protect the life, health, dignity, integrity, right to self-determination, privacy, and confidentiality of personal information of research subjects. The responsibility for the protection of research subjects must

always rest with the physician or other health care professionals and never with the research subjects, even though they have given consent.

- 10. Physicians must consider the ethical, legal and regulatory norms and standards for research involving human subjects in their own countries as well as applicable international norms and standards. No national or international ethical, legal or regulatory requirement should reduce or eliminate any of the protections for research subjects set forth in this Declaration.
- 11. Medical research should be conducted in a manner that minimises possible harm to the environment.
- 12. Medical research involving human subjects must be conducted only by individuals with the appropriate ethics and scientific education, training and qualifications. Research on patients or healthy volunteers requires the supervision of a competent and appropriately qualified physician or other health care professional.
- 13. Groups that are underrepresented in medical research should be provided appropriate access to participation in research.
- 14. Physicians who combine medical research with medical care should involve their patients in research only to the extent that this is justified by its potential preventive, diagnostic or therapeutic value and if the physician has good reason to believe that participation in the research study will not adversely affect the health of the patients who serve as research subjects.
- 15. Appropriate compensation and treatment for subjects who are harmed as a result of participating in research must be ensured.

#### Risks, Burdens and Benefits

16. In medical practice and in medical research, most interventions involve risks and burdens.

Medical research involving human subjects may only be conducted if the importance of the objective outweighs the risks and burdens to the research subjects.

17. All medical research involving human subjects must be preceded by careful assessment of predictable risks and burdens to the individuals and groups involved in the research in comparison with foreseeable benefits to them and to other individuals or groups affected by the condition under investigation.

Measures to minimise the risks must be implemented. The risks must be continuously monitored, assessed and documented by the researcher.

18. Physicians may not be involved in a research study involving human subjects unless they are confident that the risks have been adequately assessed and can be satisfactorily managed.

When the risks are found to outweigh the potential benefits or when there is conclusive proof of definitive outcomes, physicians must assess whether to continue, modify or immediately stop the study.

#### **Vulnerable Groups and Individuals**

19. Some groups and individuals are particularly vulnerable and may have an increased likelihood of being wronged or of incurring additional harm.

All vulnerable groups and individuals should receive specifically considered protection.

20. Medical research with a vulnerable group is only justified if the research is responsive to the health needs or priorities of this group and the research cannot be carried out in a non-vulnerable group. In addition, this group should stand to benefit from the knowledge, practices or interventions that result from the research.

#### Scientific Requirements and Research Protocols

- 21. Medical research involving human subjects must conform to generally accepted scientific principles, be based on a thorough knowledge of the scientific literature, other relevant sources of information, and adequate laboratory and, as appropriate, animal experimentation. The welfare of animals used for research must be respected.
- 22. The design and performance of each research study involving human subjects must be clearly described and justified in a research protocol.

The protocol should contain a statement of the ethical considerations involved and should indicate how the principles in this Declaration have been addressed. The protocol should include information regarding funding, sponsors, institutional affiliations, potential conflicts of interest, incentives for subjects and information regarding provisions for treating and/or compensating subjects who are harmed as a consequence of participation in the research study.

In clinical trials, the protocol must also describe appropriate arrangements for post-trial provisions.

#### **Research Ethics Committees**

23. The research protocol must be submitted for consideration, comment, guidance and approval to the concerned research ethics committee before the study begins. This committee must be transparent in its functioning, must be independent of the researcher, the sponsor and any other undue influence and must be duly qualified. It must take into consideration the laws and regulations of the country or countries in which the research is to be performed as well as applicable international norms and standards but these must not be allowed to reduce or eliminate any of the protections for research subjects set forth in this Declaration.

The committee must have the right to monitor ongoing studies. The researcher must provide monitoring information to the committee, especially information about any serious adverse events. No amendment to the protocol may be made without consideration and approval by the

committee. After the end of the study, the researchers must submit a final report to the committee containing a summary of the study's findings and conclusions.

## **Privacy and Confidentiality**

24. Every precaution must be taken to protect the privacy of research subjects and the confidentiality of their personal information.

#### **Informed Consent**

- 25. Participation by individuals capable of giving informed consent as subjects in medical research must be voluntary. Although it may be appropriate to consult family members or community leaders, no individual capable of giving informed consent may be enrolled in a research study unless he or she freely agrees.
- 26. In medical research involving human subjects capable of giving informed consent, each potential subject must be adequately informed of the aims, methods, sources of funding, any possible conflicts of interest, institutional affiliations of the researcher, the anticipated benefits and potential risks of the study and the discomfort it may entail, post-study provisions and any other relevant aspects of the study. The potential subject must be informed of the right to refuse to participate in the study or to withdraw consent to participate at any time without reprisal. Special attention should be given to the specific information needs of individual potential subjects as well as to the methods used to deliver the information.

After ensuring that the potential subject has understood the information, the physician or another appropriately qualified individual must then seek the potential subject's freely-given informed consent, preferably in writing. If the consent cannot be expressed in writing, the non-written consent must be formally documented and witnessed.

All medical research subjects should be given the option of being informed about the general outcome and results of the study.

- 27. When seeking informed consent for participation in a research study the physician must be particularly cautious if the potential subject is in a dependent relationship with the physician or may consent under duress. In such situations the informed consent must be sought by an appropriately qualified individual who is completely independent of this relationship.
- 28. For a potential research subject who is incapable of giving informed consent, the physician must seek informed consent from the legally authorised representative. These individuals must not be included in a research study that has no likelihood of benefit for them unless it is intended to promote the health of the group represented by the potential subject, the research cannot instead be performed with persons capable of providing informed consent, and the research entails only minimal risk and minimal burden.
- 29. When a potential research subject who is deemed incapable of giving informed consent is able to give assent to decisions about participation in research, the physician must seek that

assent in addition to the consent of the legally authorised representative. The potential subject's dissent should be respected.

- 30. Research involving subjects who are physically or mentally incapable of giving consent, for example, unconscious patients, may be done only if the physical or mental condition that prevents giving informed consent is a necessary characteristic of the research group. In such circumstances the physician must seek informed consent from the legally authorised representative. If no such representative is available and if the research cannot be delayed, the study may proceed without informed consent provided that the specific reasons for involving subjects with a condition that renders them unable to give informed consent have been stated in the research protocol and the study has been approved by a research ethics committee. Consent to remain in the research must be obtained as soon as possible from the subject or a legally authorised representative.
- 31. The physician must fully inform the patient which aspects of their care are related to the research. The refusal of a patient to participate in a study or the patient's decision to withdraw from the study must never adversely affect the patient-physician relationship.
- 32. For medical research using identifiable human material or data, such as research on material or data contained in biobanks or similar repositories, physicians must seek informed consent for its collection, storage and/or reuse. There may be exceptional situations where consent would be impossible or impracticable to obtain for such research. In such situations the research may be done only after consideration and approval of a research ethics committee.

#### Use of Placebo

33. The benefits, risks, burdens and effectiveness of a new intervention must be tested against those of the best proven intervention(s), except in the following circumstances:

Where no proven intervention exists, the use of placebo, or no intervention, is acceptable; or

Where for compelling and scientifically sound methodological reasons the use of any intervention less effective than the best proven one, the use of placebo, or no intervention is necessary to determine the efficacy or safety of an intervention

and the patients who receive any intervention less effective than the best proven one, placebo, or no intervention will not be subject to additional risks of serious or irreversible harm as a result of not receiving the best proven intervention.

Extreme care must be taken to avoid abuse of this option.

#### **Post-Trial Provisions**

34. In advance of a clinical trial, sponsors, researchers and host country governments should make provisions for post-trial access for all participants who still need an intervention identified as beneficial in the trial. This information must also be disclosed to participants during the informed consent process.

#### Research Registration and Publication and Dissemination of Results

- 35. Every research study involving human subjects must be registered in a publicly accessible database before recruitment of the first subject.
- 36. Researchers, authors, sponsors, editors and publishers all have ethical obligations with regard to the publication and dissemination of the results of research. Researchers have a duty to make publicly available the results of their research on human subjects and are accountable for the completeness and accuracy of their reports. All parties should adhere to accepted guidelines for ethical reporting. Negative and inconclusive as well as positive results must be published or otherwise made publicly available. Sources of funding, institutional affiliations and conflicts of interest must be declared in the publication. Reports of research not in accordance with the principles of this Declaration should not be accepted for publication.

#### **Unproven Interventions in Clinical Practice**

37. In the treatment of an individual patient, where proven interventions do not exist or other known interventions have been ineffective, the physician, after seeking expert advice, with informed consent from the patient or a legally authorised representative, may use an unproven intervention if in the physician's judgement it offers hope of saving life, re-establishing health or alleviating suffering. This intervention should subsequently be made the object of research, designed to evaluate its safety and efficacy. In all cases, new information must be recorded and, where appropriate, made publicly available

#### **CONTRACEPTION GUIDELINES**

The Clinical Trials Facilitation Group's recommendations related to contraception and pregnancy testing in clinical studies include the use of highly effective forms of birth control. These methods include the following:

- Combined (estrogen- and progestogen-containing) hormonal contraception associated with the inhibition of ovulation (oral, intravaginal, or transdermal)
- Progestogen-only hormonal contraception associated with the inhibition of ovulation (oral, injectable, or implantable)
- Intrauterine device (IUD)
- Intrauterine hormone-releasing system (IUS)
- Bilateral tubal occlusion
- Vasectomized male partner
  - Vasectomized partner is a highly effective birth control method provided that
    partner is the sole sexual partner of the woman of childbearing potential study
    participant and that the vasectomized partner has received medical assessment of
    the surgical success.
- Sexual abstinence (defined as refraining from heterosexual intercourse during the entire period of exposure associated with the study treatment).
  - In the context of this guidance, sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the subject.

Adapted from: Clinical Trials Facilitation Group (CTFG). Recommendations Related to Contraception and Pregnancy Testing in Clinical Trials. September 15, 2014.

Available at: https://www.hma.eu/fileadmin/dateien/Human\_Medicines/01-About\_HMA/Working\_Groups/CTFG/2014\_09\_HMA\_CTFG\_Contraception.pdf

## PROHIBITED MEDICATIONS LIST

Examples below are not exclusive.

- Any new stimulant for the treatment of ADHD that the subject was not taking at Baseline is also prohibited.
- Other medications used to treat TS are prohibited.
- Dopamine depleting medications are prohibited.
- D2 receptor antagonists are prohibited.

| Prohibited Antipsychotic Medications | |
|--------------------------------------|-----------------|
| Aripiprazole | Loxapine |
| Cisapride | Methylphenidate |
| Clonidine | Paliperidone |
| Dextroamphetamine | Pimozide |
| Dronedarone | Risperidone |
| Droperidol | Thioridazine |
| Fluoxetine | Topiramate |
| Guanfacine | Ziprasidone |
| Haloperidol | |

| Other Prohibited Medications for the Treatment of Tics | Mechanism |
|---|---|
| Any dopamine agonist (e.g., ropinire | ole, pramipexole) |
| Baclofen | GABA-B receptor agonist |
| Clonazepam | GABA-A receptor positive allosteric modulation |
| Duetetrabenazine | VMAT2 inhibitor / monoamine depleter |
| Guanfacine | Alpha-2A adrenergic receptor agonist |
| Reserpine | VMAT1/2 inhibitor / inhibits uptake of dopamine |
| Tetrabenazine | VMAT2 inhibitor / monoamine depleter |
| Valbenazine | VMAT2 inhibitor / monoamine depleter |

| Other Prohibited<br>Medications | Mechanism |
|---|---|
| Chloroethylnorapomorphine | D2 receptor antagonist |
| Chlorpromazine | D2 receptor antagonist/ antipsychotic |
| Cinnarizine | Antihistamine/ calcium channel blocker/ Interaction with D2 receptors |
| Desmethoxyfallypride | D2/D3 receptor antagonist used as PET radiotracer |
| Domperidone | D2/D3 receptor antagonist/ antiemetic |
| Eticlopride | D2 receptor antagonist |
| Fallypride | D2/D3 receptor antagonist used as PET radiotracer |
| Hydroxyzine | H1 receptor antagonist |
| Itopride | D2 receptor antagonist/used as treatment for GI disorders |
| Metclopropramide | D2 receptor antagonist/ antiemetic |

| Strong Inducers of Drug Metabolism | |
|------------------------------------|-----------------------------------|
| Apalutamide | Strong inducer of drug metabolism |
| Avasimibe | Strong inducer of drug metabolism |
| Carbamazepine | Strong inducer of drug metabolism |
| Enzalutamide | Strong inducer of drug metabolism |
| Ivosidenib | Strong inducer of drug metabolism |
| Lumacaftor | Strong inducer of drug metabolism |
| Mitotane | Strong inducer of drug metabolism |
| Phenobarbital | Strong inducer of drug metabolism |
| Phenytoin | Strong inducer of drug metabolism |
| Rifampin | Strong inducer of drug metabolism |
| Rifapentine | Strong inducer of drug metabolism |
| St John's Wort extract | Strong inducer of drug metabolism |

| The dose of Sensitive CYP? their respective labels) | 2D6 substrates that may need to be reduced (according to |
|---|---|
| Atomoxetine | Sensitive CYP2D6 substrate |
| Codeine | Sensitive CYP2D6 substrate |
| Desipramine | Sensitive CYP2D6 substrate |
| Dextromethorphan | Sensitive CYP2D6 substrate |
| Deutetrabenazine | Sensitive CYP2D6 substrate |
| Doxepin | Sensitive CYP2D6 substrate |
| Eliglustat | Sensitive CYP2D6 substrate |
| Encainide | Sensitive CYP2D6 substrate |
| Enclomiphene | Sensitive CYP2D6 substrate |
| Ibogaine | Sensitive CYP2D6 substrate |
| Metoprolol | Sensitive CYP2D6 substrate |
| Methoxyphenamine | Sensitive CYP2D6 substrate |
| Nebivolol | Sensitive CYP2D6 substrate |
| Nicergoline | Sensitive CYP2D6 substrate |
| Paroxetine | Sensitive CYP2D6 substrate |
| Perhexiline | Sensitive CYP2D6 substrate |
| Perphenazine | Sensitive CYP2D6 substrate |
| Prajmaline | Sensitive CYP2D6 substrate |
| Propafenone | Sensitive CYP2D6 substrate |
| Repinotan (IV) | Sensitive CYP2D6 substrate |
| Risperidone | Sensitive CYP2D6 substrate |
| Tamoxifen | Sensitive CYP2D6 substrate |
| Tolperisone | Sensitive CYP2D6 substrate |
| Tolterodine | Sensitive CYP2D6 substrate |
| Tramadol | Sensitive CYP2D6 substrate |
| Traxoprodil | Sensitive CYP2D6 substrate |
| Trimipramine | Sensitive CYP2D6 substrate |
| Tropisetron | Sensitive CYP2D6 substrate |
| Venlafaxine | Sensitive CYP2D6 substrate |
| Vernakalant | Sensitive CYP2D6 substrate |

| OATP1B1 substrates: dose of these OATP1B1 substrates should be adjusted based on their label | |
|---|---|
| Bosentan | OATP1B1 substrate |
| Cerivastatin (acid) | OATP1B1 substrate |
| Clazosentan | OATP1B1 substrate |
| Danoprevir | OATP1B1 substrate |
| Eluxadoline | OATP1B1 substrate |
| Fimasartan | OATP1B1 substrate |
| Fluvastatin | OATP1B1 substrate |
| Glecaprevir | OATP1B1 substrate |
| Letermovir | OATP1B1 substrate |
| Pitavastatin (acid) | OATP1B1 substrate |
| Rosuvastatin (acid) | OATP1B1 substrate |
| Velpatasvir | OATP1B1 substrate |
| Voxilaprevir | OATP1B1 substrate |

| PGP substrates: dose of these PGP substrates should be adjusted based on their respective labels | |
|---|---|
| Acalabrutinib | PGP substrates |
| Adafosbuvir (AL-335) | PGP substrates |
| Albendazole | PGP substrates |
| Aliskiren | PGP substrates |
| Alisporivir | PGP substrates |
| Ambrisentan | PGP substrates |
| Amd070 | PGP substrates |
| Amenamevir | PGP substrates |
| Apixaban | PGP substrates |
| Asunaprevir | PGP substrates |
| Atecegatran metoxil | PGP substrates |
| Atorvastatin (acid) | PGP substrates |
| Avatrombopag | PGP substrates |
| Azithromycin | PGP substrates |
| Betrixaban | PGP substrates |
| Bictegravir | PGP substrates |
| Buprenorphine | PGP substrates |

| Celiprolol | PGP substrates |
|---------------------|----------------|
| Cerivastatin (acid) | PGP substrates |
| Colchicine | PGP substrates |
| Copanlisib | PGP substrates |
| Cp-481,715 | PGP substrates |
| Cyclosporine | PGP substrates |
| Dabigatran | PGP substrates |
| Danoprevir | PGP substrates |
| Deflazacort | PGP substrates |
| Dicloxacillin | PGP substrates |
| Digoxin | PGP substrates |
| Docetaxel | PGP substrates |
| Domperidone | PGP substrates |
| Doravirine | PGP substrates |
| Doxorubicin | PGP substrates |
| Edoxaban | PGP substrates |
| Elbasvir | PGP substrates |
| Emtricitabine | PGP substrates |
| Erlotinib | PGP substrates |
| Erythromycin | PGP substrates |
| Etoposide | PGP substrates |
| Everolimus | PGP substrates |
| Fentanyl | PGP substrates |
| Fexofenadine | PGP substrates |
| Glecaprevir | PGP substrates |
| Idarubicin | PGP substrates |
| Indinavir | PGP substrates |
| Irinotecan | PGP substrates |
| Itraconazole | PGP substrates |
| Ivosidenib | PGP substrates |
| Lapatinib | PGP substrates |
| Larotrectinib | PGP substrates |
| Ledipasvir | PGP substrates |

| PGP substrates: dose of based on their respective | these PGP substrates should be adjusted e labels |
|---|---|
| Letermovir | PGP substrates |
| Linezolid | PGP substrates |
| Loperamide | PGP substrates |
| Losartan | PGP substrates |
| Maraviroc | PGP substrates |
| Maraviroc | PGP substrates |
| Mirabegron | PGP substrates |
| Mitoxantrone | PGP substrates |
| Morphine | PGP substrates |
| Nadolol | PGP substrates |
| Naldemedine | PGP substrates |
| Naloxegol | PGP substrates |
| Nevirapine | PGP substrates |
| Nintedanib | PGP substrates |
| Octreotide | PGP substrates |
| Olodaterol | PGP substrates |
| Paclitaxel | PGP substrates |
| Paritaprevir | PGP substrates |
| Paroxetine | PGP substrates |
| Pazopanib | PGP substrates |
| Phenytoin | PGP substrates |
| Pibrentasvir | PGP substrates |
| Pravastatin (acid) | PGP substrates |
| Proguanil | PGP substrates |
| Quetiapine | PGP substrates |
| Quinidine | PGP substrates |
| Ranitidine | PGP substrates |
| Ranolazine | PGP substrates |
| Rivaroxaban | PGP substrates |
| Rosuvastatin (acid) | PGP substrates |
| Saquinavir | PGP substrates |
| Selexipag | PGP substrates |
| Simeprevir | PGP substrates |

| PGP substrates: dose of these PGP substrates should be adjusted based on their respective labels | |
|---|---|
| Simvastatin (lactone) | PGP substrates |
| Sirolimus | PGP substrates |
| Sofosbuvir | PGP substrates |
| Sotrastaurin | PGP substrates |
| Tacrolimus | PGP substrates |
| Talinolol | PGP substrates |
| Tedisamil | PGP substrates |
| Teneligliptin | PGP substrates |
| Tenofovir | PGP substrates |
| Ticagrelor | PGP substrates |
| Velpatasvir | PGP substrates |
| Venetoclax | PGP substrates |
| Venlafaxine | PGP substrates |
| Verapamil | PGP substrates |
| Vinblastine | PGP substrates |
| Vincristine | PGP substrates |
| Voclosporin | PGP substrates |
| Ximelagatran | PGP substrates |

| UGT1A1 substrates: dose of these UGT1A1 substrates should be adjusted based on their respective labels | |
|---|---|
| Clopidogrel | UGT1A9 substrate |
| Furosemide | UGT1A9 substrate |
| Mycophenolic acid | UGT1A9 substrate |
| Probenecid | UGT1A9 substrate |
| Propofol | UGT1A9 substrate |